CLINICAL TRIAL: NCT01421069
Title: AN OPEN-LABEL EXTENSION STUDY TO ASSESS THE LONG-TERM SAFETY AND CLINICAL BENEFIT OF ETANERCEPT IN CHILDREN AND ADOLESCENTS WITH EXTENDED OLIGOARTICULAR JUVENILE IDIOPATHIC ARTHRITIS, ENTHESITIS-RELATED ARTHRITIS, OR PSORIATIC ARTHRITIS WHO WERE PREVIOUSLY ENROLLED IN PROTOCOL 0881A1-3338-WW(B1801014)
Brief Title: Extension Study Evaluating Etanercept in 3 Subtypes of Childhood Arthritis
Acronym: CLIPPER2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: B1801023; 0881A1-3342 (Other: Alias Study Number); 2010-023802-10 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-04

CONDITIONS: Juvenile Idiopahtic Arthritis
Keywords: Use of etanercept to treat pediatric subjects with extended oligoarticular JIA; enthestitis related arthritis (ERA); or psoriatic arthritis (PsA).
MeSH Terms: conditions — Arthritis, Psoriatic; Salivary Gland Adenoma, Pleomorphic | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Subjects aged <18 years and less than or equal to 62 kg will receive etanercept SC at a dose of 0.8 mg/kg QW (up to a maximum dose of 50 mg QW).
  Subjects aged greater than or equal to 18 years or >62 kg will receive etanercept SC at a dose of 50 mg QW.

SUMMARY:
This is a 8-year extension study in pediatric subjects who have been diagnosed with one of 3 subtypes of Juvenile Idiopathic Arthritis (JIA) [extended oligoarticular JIA, enthestitis related arthritis (ERA), or psoriatic arthritis (PsA)] who have completed approximately 96 weeks of participation in study 0881A1-3338 (B1801014). The study contains an active treatment period, withdrawal/re-treatment period and a observational period (non-treatment).

ELIGIBILITY:
Inclusion Criteria:

Receipt of at least 1 dose of investigational product (etanercept) and participation for approximately 96 weeks in study 0881A1-3338 (B1801014)

Personally signed and dated informed consent document (and assent document, as applicable) indicating the subject (or legally representative/guardian) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

Exclusion criteria for subject planning to continue investigational product:

withdrawal from investigational product in study 0881A1-3338 for any reason (safety or non-safety).

History of maliginancy other than squamous cell, basal cell carcinoma or cervical carcinoma in situ.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, Sydney, New South Wales
  - Royal Children's Hospital, Parkville, Melbourne, Victoria
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Servimed S.A.S, Bucaramanga, Santander Department, Colombia
- Czechia (3):
  - Fakultni nemocnice Brno - Detska nemocnice, Ambulance detske revmatologie, Brno
  - Klinika detskeho a dorostoveho lekarstvi 1. LF UK a VFN v Praze, Prague
  - Revmatologicky ustav, Prague
- France (2):
  - Hopital Cochin, Paris
  - Hopital NECKER-Enfants Malades, Paris
- Germany (4):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Schön Klinik Hamburg Eilbek, Hamburg
  - Asklepios Klinik Sankt Augustin GmbH, Zentrum fuer Kinder- und Jugendrheumatologie, Saint Augustin
- Semmelweis Egyetem, Budapest, Hungary
- Centro di Ricerca Clinica - Fondazione dell'Universita' degli Studi "G. D'Annunzio", Chieti Scalo, Italy
- Latvia (2):
  - University Children Hospital Gailezers, Riga
  - University Children Hospital, Riga
- Children's Hospital at Vilnius University Hospital "Santaros klinikos", Vilnius, Lithuania
- CLIDITER S.A. de C.V., México, D.F., Mexico
- Universitair Ziekenhuis Utrecht, Wilhelmina Kinderziekenhuis, Room number KC 03-063, Utrecht, Netherlands
- Depart. of Rheumatology, Oslo, Norway
- Poland (4):
  - Wojewodzki Szpital Dzieciecy im. J. Brudzinskiego, Bydgoszcz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie,, Krakow
  - Instytut Reumatologii im. prof. dr hab. med. Eleonory Reicher, Klinika i, Warsaw
  - Szpital Specjalistyczny im. A. Falkiewicza we Wroclawiu, Oddzial Pediatryczno - Reumatologiczny, Wroclaw
- Russia (2):
  - FGBNU Research Institute of Rheumatology n.a. V.A. Nasonovoy, Moscow
  - SBEI HPE Saint Petersburg State Pediatric Medical University, Saint Petersburg
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Children's Clinic of Internal Medicine, Niš
- Narodny ustav reumatickych chorob, Piešťany, Slovakia
- University Medical Centre Ljubljana, University Children's Hospital, Ljubljana, Slovenia
- Spain (3):
  - Hospital San Juan de Dios, Esplugues de Llobregat, Barcelona
  - Hospital Universitario RamÃ³n y Cajal, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vojinovic J, Foeldvari I, Dehoorne J, Panaviene V, Susic G, Horneff G, Stanevicha V, Kobusinska K, Zuber Z, Dobrzyniecka B, Akikusa J, Avcin T, Borlenghi C, Arthur E, Tatulych SY, Zang C, Tsekouras V, Vlahos B, Martini A, Ruperto N. Ten-year safety and clinical benefit from open-label etanercept treatment in children and young adults with juvenile idiopathic arthritis. Rheumatology (Oxford). 2024 Jan 4;63(1):140-148. doi: 10.1093/rheumatology/kead183. PMID 37140539
- [Derived] Foeldvari I, Constantin T, Vojinovic J, Horneff G, Chasnyk V, Dehoorne J, Panaviene V, Susic G, Stanevicha V, Kobusinska K, Zuber Z, Dobrzyniecka B, Nikishina I, Bader-Meunier B, Breda L, Dolezalova P, Job-Deslandre C, Rumba-Rozenfelde I, Wulffraat N, Pedersen RD, Bukowski JF, Vlahos B, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). Etanercept treatment for extended oligoarticular juvenile idiopathic arthritis, enthesitis-related arthritis, or psoriatic arthritis: 6-year efficacy and safety data from an open-label trial. Arthritis Res Ther. 2019 May 23;21(1):125. doi: 10.1186/s13075-019-1916-9. PMID 31122296
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801023&StudyName=Extension%20Study%20Evaluating%20Etanercept%20in%203%20Subtypes%20of%20Childhood%20Arthritis%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an extension study in pediatric participants diagnosed with one of three subtypes of juvenile idiopathic arthritis (JIA): extended oligoarticular JIA, enthesitis related arthritis (ERA), or psoriatic arthritis (PsA) and had received at least one dose of Etanercept and completed approximately 96 weeks of participation in study B1801014 (NCT00962741).
Pre-assignment Details: Total 127 participants were enrolled and treated in parent study, B1801014 (NCT00962741) and included in analysis of this extension study. Total 109 participants from the Parent study were enrolled in this extension study, B1801023. Out of which 10 participants directly entered into observational phase and did not receive treatment in this extension study. The extension study has 3 periods: active treatment period, withdrawal/re-treatment period and observational period.
Groups:
- Etanercept: Participants who completed 96 weeks of Etanercept treatment in study B1801014 and eligible to continue Etanercept in study B1801023, entered directly into active treatment period to receive Etanercept subcutaneous dose of 0.8 milligram/kilogram once a week, for maximum of 96 months. Eligible participants from active treatment, who either met Wallace definition for clinically inactive disease for at least 6 months or had good clinical response and would benefit from treatment withdrawal entered withdrawal period. Eligible participants requiring re-treatment per investigator's judgment entered re-treatment period. Participants who discontinued treatment prior to 96 weeks in study B1801014 or not eligible to continue treatment in B1801023 entered directly into observational period. Participants who discontinued treatment/study period, prior to completion also entered into observational period. In observational period, all participants were followed up for maximum of 96 months from time of initial entry into this study.
Period: Parent Study
Arm/Group | Etanercept
Started | 127
Completed | 119
Not Completed | 8
Not completed — drug ineffective+prohibited drug taken | 1
Not completed — Failed to return | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1
Period: Overall Period for Extension Study
Arm/Group | Etanercept
Started | 109
Enrolled Into Active Treatment Period | 99
Enrolled Into Observational Period | 10
Completed | 84 (27 participants completed study in Active Treatment period, 45 completed study in Observational Period, 5 completed study in Re-treatment Period, and 7 completed study in Withdrawal Period.)
Not Completed | 25
Not completed — Other | 2
Not completed — Medication error without associated adverse event | 1
Not completed — No longer willing to participate | 14
Not completed — Pregnancy | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 1
Period: Active Treatment Period
Arm/Group | Etanercept
Started | 99
ERA | 31
PsA | 23
Completed | 27
Not Completed | 72
Not completed — Other | 1
Not completed — No longer willing to participate in study | 8
Not completed — Insufficient clinical response | 1
Not completed — Medication error without associated adverse event | 1
Not completed — Pregnancy | 1
Not completed — Adverse Event | 1
Not completed — Enrolled in withdrawal period | 30
Not completed — Enrolled in observational period | 29
Period: 2a. Withdrawal Period
Arm/Group | Etanercept
Started | 30 (Participants from active treatment, who either met Wallace definition for clinically inactive disease for at least 6 months or had good clinical response and would benefit from treatment withdrawal entered withdrawal period.)
ERA | 9
PsA | 5
Completed | 7
Not Completed | 23
Not completed — No longer willing to participate in study | 2
Not completed — Lost to Follow-up | 1
Not completed — Enrolled in observational period | 7
Not completed — Enrolled in re-treatment period | 13
Period: 2b. Retreatment Period
Arm/Group | Etanercept
Started | 13 (Participants requiring re-treatment per investigator's judgment entered re-treatment period.)
ERA | 2
PsA | 3
Completed | 5
Not Completed | 8
Not completed — Enrolled in observational period | 7
Not completed — Protocol Violation | 1
Period: Observational Period
Arm/Group | Etanercept
Started | 53 (10 participants entered directly from Parent study B1801014 (NCT00962741))
Completed | 45
Not Completed | 8
Not completed — Other | 1
Not completed — No longer willing to participate in study | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants from parent study B1801014 (NCT00962741) who received at least 1 dose of investigational product in parent study, regardless of whether they received any investigational product during the extension study.
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.28 (4.49) [lower limit 4.49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 101
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Malignancy: All Periods of Parent and Extension Study
Description: Number of participants who had adverse event (AE) of malignancy were reported. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: First dose of study medication in parent study up to 96 months in the extension study, for a maximum duration of 118 months (22 months of parent study and 96 months of extension study)
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 1

2. Secondary Outcome: Number of Participants With Serious Adverse Events: All Periods of Parent and Extension Study
Description: A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: as for outcome 1
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 45

3. Secondary Outcome: Number of Participants With Serious Infections: All Periods of Parent and Extension Study
Description: Serious infections were defined as any infections those were life threatening or resulted in disability, infections requiring intravenous antibiotic treatment and hospitalization.
Time Frame: as for outcome 1
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 14

4. Secondary Outcome: Number of Participants With Medically Important Infections: All Periods of Parent and Extension Study
Description: Medically important infections were defined as an infection requiring parenteral (intravenous [IV], intramuscular [IM]) anti-infective agent(s) and/or hospitalization.
Time Frame: as for outcome 1
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 12

5. Secondary Outcome: Number of Participants With Infections: All Periods of Parent and Extension Study
Description: Number of participants who had infections as AEs were reported. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: as for outcome 1
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 111

6. Secondary Outcome: Number of Participants With Treatment Emergent Infections and Injection Site Reactions: All Periods of Extension Study
Description: Number of participants who had treatment emergent infections and injection site reactions as adverse events were reported. Treatment emergent infections were infections occurring in a participant who received study medication without regard to possibility of causal relationship to it. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: Extension study: Baseline (Day 1) up to 30 days after the last dose of investigational product (maximum up to 97 months)
Population: Analysis population included all participants who were enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants
  Treatment emergent infections | 67
  Injection site reactions | 6

7. Secondary Outcome: Number of Participants With Infections: Extension Study: Withdrawal Period
Description: Number of participants who had treatment emergent infections as AEs were reported. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: Extension study: Day of study treatment withdrawal up to entering re-treatment period or observational period (for a maximum of 96 months)
Population: Withdrawal analysis set (WAS) included those participants who entered the withdrawal period.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Participants
  Infections | 8
  Infections considered preventable by vaccination | 1

8. Secondary Outcome: Number of Participants Withdrawn Due to Adverse Events: All Periods of Parent and Extension Study
Description: Participants withdrew from the study due to AEs were reported. An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Time Frame: as for outcome 1
Population: Analysis population included all participants who were enrolled in the parent and extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants
  Due to infections | 3
  Due to other adverse events | 14

9. Secondary Outcome: Number of Participants Withdrawn Due to Adverse Events: Extension Study: Withdrawal Period
Description: as for outcome 8
Time Frame: as for outcome 7
Population: WAS included those participants who entered the withdrawal period.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Participants | 0

10. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Laboratory Abnormalities Based on National Cancer Institute Criteria Version 4.03: All Periods of Extension Study
Description: Abnormality of laboratory parameters was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: as for outcome 6
Population: Analysis population included all participants who were enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants
  Grade 3 | 2
  Grade 4 | 0

11. Secondary Outcome: Change From Baseline of Parent Study in Z-Score at Month 12, 24, 36, 48, 60, 72, 84 and 96 of Extension Study: Active Treatment Period
Description: Growth parameters including weight, height and body-mass index (BMI) were compared to the standard growth data by using Z-Score. Z-Score is a statistical measure to evaluate how a single data point or mean compares to a standard. A Z-Score describes whether a mean is above or below the standard and how unusual the measurement is. Z-scores range from -3 to +3. A Z-score of 0 indicates the same mean, greater than (>) 0 a greater mean, and less than (<0) a lesser mean than the standard.
Time Frame: Baseline of the parent study; Month 12, 24, 36, 48, 60, 72, 84 and 96 active treatment period of extension study
Population: FAS included all participants in the parent study who received at least 1 dose of investigational product regardless of whether they received any investigational product during the extension study. Here, "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 99
z-score
  Change at Month 12 of extension study: Height: number analyzed (Participants) | 88
  Change at Month 12 of extension study: Height | 0.22 (0.46)
  Change at Month 24 of extension study: Height: number analyzed (Participants) | 55
  Change at Month 24 of extension study: Height | 0.17 (0.56)
  Change at Month 36 of extension study: Height: number analyzed (Participants) | 43
  Change at Month 36 of extension study: Height | 0.21 (0.66)
  Change at Month 48 of extension study: Height: number analyzed (Participants) | 28
  Change at Month 48 of extension study: Height | 0.19 (0.58)
  Change at Month 60 of extension study: Height: number analyzed (Participants) | 13
  Change at Month 60 of extension study: Height | 0.25 (0.67)
  Change at Month 72 of extension study: Height: number analyzed (Participants) | 10
  Change at Month 72 of extension study: Height | 0.30 (0.90)
  Change at Month 84 of extension study: Height: number analyzed (Participants) | 5
  Change at Month 84 of extension study: Height | 0.09 (0.53)
  Change at Month 96 of extension study: Height: number analyzed (Participants) | 4
  Change at Month 96 of extension study: Height | 0.16 (0.63)
  Change at Month 12 of extension study: Weight: number analyzed (Participants) | 81
  Change at Month 12 of extension study: Weight | 0.05 (0.60)
  Change at Month 24 of extension study: Weight: number analyzed (Participants) | 53
  Change at Month 24 of extension study: Weight | -0.04 (0.68)
  Change at Month 36 of extension study: Weight: number analyzed (Participants) | 40
  Change at Month 36 of extension study: Weight | -0.06 (0.72)
  Change at Month 48 of extension study: Weight: number analyzed (Participants) | 25
  Change at Month 48 of extension study: Weight | -0.00 (0.71)
  Change at Month 60 of extension study: Weight: number analyzed (Participants) | 13
  Change at Month 60 of extension study: Weight | 0.25 (0.64)
  Change at Month 72 of extension study: Weight: number analyzed (Participants) | 10
  Change at Month 72 of extension study: Weight | 0.45 (0.74)
  Change at Month 84 of extension study: Weight: number analyzed (Participants) | 5
  Change at Month 84 of extension study: Weight | 0.04 (0.62)
  Change at Month 96 of extension study: Weight: number analyzed (Participants) | 4
  Change at Month 96 of extension study: Weight | 0.27 (0.68)
  Change at Month 12 of extension study: BMI: number analyzed (Participants) | 88
  Change at Month 12 of extension study: BMI | -0.03 (0.77)
  Change at Month 24 of extension study: BMI: number analyzed (Participants) | 55
  Change at Month 24 of extension study: BMI | -0.13 (0.86)
  Change at Month 36 of extension study: BMI: number analyzed (Participants) | 43
  Change at Month 36 of extension study: BMI | -0.19 (0.79)
  Change at Month 48 of extension study: BMI: number analyzed (Participants) | 28
  Change at Month 48 of extension study: BMI | -0.17 (0.87)
  Change at Month 60 of extension study: BMI: number analyzed (Participants) | 13
  Change at Month 60 of extension study: BMI | 0.02 (0.86)
  Change at Month 72 of extension study: BMI: number analyzed (Participants) | 10
  Change at Month 72 of extension study: BMI | 0.26 (1.00)
  Change at Month 84 of extension study: BMI: number analyzed (Participants) | 5
  Change at Month 84 of extension study: BMI | 0.00 (0.99)
  Change at Month 96 of extension study: BMI: number analyzed (Participants) | 4
  Change at Month 96 of extension study: BMI | 0.27 (1.21)

12. Secondary Outcome: Change From Baseline in Z-Score at Month 12, 24, 36, 42, 48, 60, 72, 84 and 96 of Extension Study: Withdrawal Period
Description: Growth parameters including weight, height and BMI were compared to the standard growth data by using Z-Score. Z-Score is a statistical measure to evaluate how a single data point or mean compares to a standard. A Z-Score describes whether a mean is above or below the standard and how unusual the measurement is. Z-scores range from -3 to +3. A Z-score of 0 indicates the same mean, >0 a greater mean, and <0 a lesser mean than the standard.
Time Frame: Baseline of the extension study; Month 12, 24, 36, 42, 48, 60, 72, 84 and 96 withdrawal period of extension study
Population: WAS included participants who entered the withdrawal period. Here, "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 30
z-score
  Change at Month 12: Height: number analyzed (Participants) | 9
  Change at Month 12: Height | -0.10 (0.21)
  Change at Month 24: Height: number analyzed (Participants) | 5
  Change at Month 24: Height | -0.13 (0.28)
  Change at Month 36: Height: number analyzed (Participants) | 3
  Change at Month 36: Height | 0.03 (0.05)
  Change at Month 42: Height: number analyzed (Participants) | 0
  Change at Month 48: Height: number analyzed (Participants) | 1
  Change at Month 48: Height | 0.26
  Change at Month 60: Height: number analyzed (Participants) | 1
  Change at Month 60: Height | 0.41
  Change at Month 72: Height: number analyzed (Participants) | 1
  Change at Month 72: Height | 0.52
  Change at Month 84: Height: number analyzed (Participants) | 0
  Change at Month 96: Height: number analyzed (Participants) | 0
  Change at Month 12: Weight: number analyzed (Participants) | 9
  Change at Month 12: Weight | -0.07 (0.25)
  Change at Month 24: Weight: number analyzed (Participants) | 4
  Change at Month 24: Weight | -0.09 (0.35)
  Change at Month 36: Weight: number analyzed (Participants) | 3
  Change at Month 36: Weight | -0.05 (0.42)
  Change at Month 42: Weight: number analyzed (Participants) | 3
  Change at Month 42: Weight | -0.47 (1.08)
  Change at Month 48: Weight: number analyzed (Participants) | 1
  Change at Month 48: Weight | 0.22
  Change at Month 60: Weight: number analyzed (Participants) | 1
  Change at Month 60: Weight | 0.46
  Change at Month 72: Weight: number analyzed (Participants) | 1
  Change at Month 72: Weight | 0.60
  Change at Month 84: Weight: number analyzed (Participants) | 0
  Change at Month 96: Weight: number analyzed (Participants) | 0
  Change at Month 12: BMI: number analyzed (Participants) | 9
  Change at Month 12: BMI | -0.04 (0.24)
  Change at Month 24: BMI: number analyzed (Participants) | 5
  Change at Month 24: BMI | -0.14 (0.30)
  Change at Month 36: BMI: number analyzed (Participants) | 3
  Change at Month 36: BMI | 0.06 (0.51)
  Change at Month 42: BMI: number analyzed (Participants) | 0
  Change at Month 48: BMI: number analyzed (Participants) | 1
  Change at Month 48: BMI | 0.51
  Change at Month 60: BMI: number analyzed (Participants) | 1
  Change at Month 60: BMI | 0.72
  Change at Month 72: BMI: number analyzed (Participants) | 1
  Change at Month 72: BMI | 0.72
  Change at Month 84: BMI: number analyzed (Participants) | 0
  Change at Month 96: BMI: number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in Z-Score at Month 12, 24, 36, 42, 48, 60, 72, 84 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 12
Time Frame: Baseline of the extension study; Month 12, 24, 36, 42, 48, 60, 72, 84 and 96 re-treatment period of extension study
Population: Re-treatment analysis set (RTAS) included those participants who entered the re-treatment period. Here, "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 13
z-score
  Change at Month 12: Height: number analyzed (Participants) | 9
  Change at Month 12: Height | -0.21 (0.31)
  Change at Month 24: Height: number analyzed (Participants) | 8
  Change at Month 24: Height | -0.19 (0.43)
  Change at Month 36: Height: number analyzed (Participants) | 6
  Change at Month 36: Height | -0.19 (0.41)
  Change at Month 42: Height: number analyzed (Participants) | 0
  Change at Month 48: Height: number analyzed (Participants) | 4
  Change at Month 48: Height | 0.07 (0.12)
  Change at Month 60: Height: number analyzed (Participants) | 2
  Change at Month 60: Height | -0.08 (0.27)
  Change at Month 72: Height: number analyzed (Participants) | 0
  Change at Month 84 Height: number analyzed (Participants) | 0
  Change at Month 96: Height: number analyzed (Participants) | 0
  Change at Month 12: Weight: number analyzed (Participants) | 9
  Change at Month 12: Weight | 0.08 (0.26)
  Change at Month 24: Weight: number analyzed (Participants) | 8
  Change at Month 24: Weight | -0.07 (0.32)
  Change at Month 36: Weight: number analyzed (Participants) | 7
  Change at Month 36: Weight | -0.15 (0.43)
  Change at Month 42: Weight: number analyzed (Participants) | 5
  Change at Month 42: Weight | -0.36 (0.42)
  Change at Month 48: Weight: number analyzed (Participants) | 4
  Change at Month 48: Weight | -0.33 (0.58)
  Change at Month 60: Weight: number analyzed (Participants) | 2
  Change at Month 60: Weight | -0.57 (0.12)
  Change at Month 72: Weight: number analyzed (Participants) | 1
  Change at Month 72: Weight | -1.06
  Change at Month 84: Weight: number analyzed (Participants) | 0
  Change at Month 96: Weight: number analyzed (Participants) | 0
  Change at Month 12: BMI: number analyzed (Participants) | 9
  Change at Month 12: BMI | 0.27 (0.60)
  Change at Month 24: BMI: number analyzed (Participants) | 8
  Change at Month 24: BMI | 0.01 (0.71)
  Change at Month 36: BMI: number analyzed (Participants) | 6
  Change at Month 36: BMI | -0.17 (0.83)
  Change at Month 42: BMI: number analyzed (Participants) | 0
  Change at Month 48: BMI: number analyzed (Participants) | 4
  Change at Month 48: BMI | -0.59 (0.90)
  Change at Month 60: BMI: number analyzed (Participants) | 2
  Change at Month 60: BMI | -0.85 (0.16)
  Change at Month 72: BMI: number analyzed (Participants) | 0
  Change at Month 84: BMI: number analyzed (Participants) | 0
  Change at Month 96: BMI: number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline (of Parent Study) in Tanner Assessment Score for Participants Aged <18 Years at Month 12, 24, 36, 48, 60, 72, 84 and 96 of Extension Study: Active Treatment Period
Description: Tanner assessment score: used to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; male pubertal development staged by size of the genitalia and development of pubic hair. Tanner assessment score ranged from 1 (no development) to 5 (adult-like development in quantity and size), higher scores indicated more development.
Time Frame: Baseline of the parent study; Month 12, 24, 36, 48, 60, 72, 84 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on a scale
  Change at Month 12 of extension study: number analyzed (Participants) | 89
  Change at Month 12 of extension study | 0.78 (0.88)
  Change at Month 24 of extension study: number analyzed (Participants) | 61
  Change at Month 24 of extension study | 1.02 (0.99)
  Change at Month 36 of extension study: number analyzed (Participants) | 53
  Change at Month 36 of extension study | 1.35 (1.19)
  Change at Month 48 of extension study: number analyzed (Participants) | 40
  Change at Month 48 of extension study | 1.69 (1.36)
  Change at Month 60 of extension study: number analyzed (Participants) | 14
  Change at Month 60 of extension study | 1.70 (1.44)
  Change at Month 72 of extension study: number analyzed (Participants) | 4
  Change at Month 72 of extension study | 2.25 (1.50)
  Change at Month 84 of extension study: number analyzed (Participants) | 2
  Change at Month 84 of extension study | 3.00 (1.41)
  Change at Month 96 of extension study: number analyzed (Participants) | 1
  Change at Month 96 of extension study | 4.00

15. Secondary Outcome: Change From Baseline in Tanner Assessment Score for Participants Aged <18 Years at Month 12, 24, 36, 48, 60, 72, 84 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 14
Time Frame: Baseline of the extension study; Month 12, 24, 36, 48, 60, 72, 84 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on a scale
  Change at Month 12: number analyzed (Participants) | 6
  Change at Month 12 | 0.08 (0.20)
  Change at Month 24: number analyzed (Participants) | 4
  Change at Month 24 | 0.38 (0.75)
  Change at Month 36: number analyzed (Participants) | 1
  Change at Month 36 | 0.00
  Change at Month 48: number analyzed (Participants) | 2
  Change at Month 48 | 0.00 (0.00)
  Change at Month 60: number analyzed (Participants) | 1
  Change at Month 60 | 0.00
  Change at Month 72: number analyzed (Participants) | 1
  Change at Month 72 | 0.00
  Change at Month 84: number analyzed (Participants) | 0
  Change at Month 96: number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline in Tanner Assessment Score for Participants Aged <18 Years at Month 12, 24, 36, 48, 60, 72, 84 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 14
Time Frame: Baseline of the extension study; Month 12, 24, 36, 48, 60, 72, 84 and 96 re-treatment period of extension study
Population: RTAS included those participants who entered the re-treatment period. Here, "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on a scale
  Change at Month 12: number analyzed (Participants) | 9
  Change at Month 12 | 0.04 (0.11)
  Change at Month 24: number analyzed (Participants) | 9
  Change at Month 24 | 0.52 (0.75)
  Change at Month 36: number analyzed (Participants) | 7
  Change at Month 36 | 1.52 (1.73)
  Change at Month 48: number analyzed (Participants) | 5
  Change at Month 48 | 1.27 (1.64)
  Change at Month 60: number analyzed (Participants) | 1
  Change at Month 60 | 1.67
  Change at Month 72: number analyzed (Participants) | 0
  Change at Month 84: number analyzed (Participants) | 0
  Change at Month 96: number analyzed (Participants) | 0

17. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 30% (ACR30) Pediatric Response (ACR30PR) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96 of Extension Study: Active Treatment Period
Description: ACR30PR: >=30% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria: physician's global assessment (on 21-circle VAS ranging 0 [no disease activity] to 10 [maximum disease activity],higher score=more severe disease), patient global assessment (on 21-circle VAS ranging 0 [very well] to 10 [very poor],higher score=higher pain), childhood health assessment questionnaire ([CHAQ] Participants >18 years assessed for functional disability, discomfort. Ability to dressing, arising, eat, walk, hygiene, reach, grip, common activities were distributed in 30 items. Each item scored from 0 [no difficulty] to 3 [unable to do]. Highest score for each domain was score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered and ranged from 0 [no difficulty] to 3 [extreme difficulty], where higher scores=more functional disability and discomfort), number of active joints and joints with limited range of motion, C-reactive protein.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 23
  Month 6 | 95.7 [78.1 to 99.9]
  Month 12: number analyzed (Participants) | 61
  Month 12 | 98.4 [91.2 to 100]
  Month 18: number analyzed (Participants) | 61
  Month 18 | 96.7 [88.7 to 99.6]
  Month 24: number analyzed (Participants) | 55
  Month 24 | 100 [93.5 to 100]
  Month 30: number analyzed (Participants) | 53
  Month 30 | 100 [93.3 to 100]
  Month 36: number analyzed (Participants) | 48
  Month 36 | 100 [92.6 to 100]
  Month 42: number analyzed (Participants) | 46
  Month 42 | 95.7 [85.2 to 99.5]
  Month 48: number analyzed (Participants) | 43
  Month 48 | 97.7 [87.7 to 99.9]
  Month 54: number analyzed (Participants) | 38
  Month 54 | 100 [90.7 to 100]
  Month 60: number analyzed (Participants) | 34
  Month 60 | 100 [89.7 to 100]
  Month 66: number analyzed (Participants) | 31
  Month 66 | 100 [88.8 to 100]
  Month 72: number analyzed (Participants) | 25
  Month 72 | 100 [86.3 to 100]
  Month 78: number analyzed (Participants) | 24
  Month 78 | 100 [85.8 to 100]
  Month 84: number analyzed (Participants) | 21
  Month 84 | 100 [83.9 to 100]
  Month 90: number analyzed (Participants) | 22
  Month 90 | 100 [84.6 to 100]
  Month 96: number analyzed (Participants) | 16
  Month 96 | 100 [79.4 to 100]

18. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 30% (ACR30) Pediatric Response (ACR30PR) at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 17
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 23
  Month 1 | 95.7 [78.1 to 99.9]
  Month 3: number analyzed (Participants) | 15
  Month 3 | 100 [78.2 to 100]
  Month 6: number analyzed (Participants) | 11
  Month 6 | 100 [71.5 to 100]
  Month 9: number analyzed (Participants) | 9
  Month 9 | 88.9 [51.8 to 99.7]
  Month 12: number analyzed (Participants) | 9
  Month 12 | 88.9 [51.8 to 99.7]
  Month 18: number analyzed (Participants) | 8
  Month 18 | 100 [63.1 to 100]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 100 [47.8 to 100]
  Month 30: number analyzed (Participants) | 4
  Month 30 | 100 [39.8 to 100]
  Month 36: number analyzed (Participants) | 4
  Month 36 | 100 [39.8 to 100]
  Month 42: number analyzed (Participants) | 4
  Month 42 | 100 [39.8 to 100]
  Month 48: number analyzed (Participants) | 3
  Month 48 | 66.7 [9.4 to 99.2]
  Month 54: number analyzed (Participants) | 1
  Month 54 | 100 [2.5 to 100]
  Month 60: number analyzed (Participants) | 2
  Month 60 | 100 [15.8 to 100]
  Month 66: number analyzed (Participants) | 1
  Month 66 | 100 [2.5 to 100]
  Month 72: number analyzed (Participants) | 1
  Month 72 | 100 [2.5 to 100]
  Month 78: number analyzed (Participants) | 0
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

19. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 30% (ACR30) Pediatric Response (ACR30PR) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Re-treatment Period:
Description: as for outcome 17
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3: number analyzed (Participants) | 12
  Month 3 | 100 [73.5 to 100]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 100 [73.5 to 100]
  Month 9: number analyzed (Participants) | 12
  Month 9 | 91.7 [61.5 to 99.8]
  Month 12: number analyzed (Participants) | 11
  Month 12 | 90.9 [58.7 to 99.8]
  Month 18: number analyzed (Participants) | 10
  Month 18 | 100 [69.2 to 100]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 100 [63.1 to 100]
  Month 30: number analyzed (Participants) | 9
  Month 30 | 100 [66.4 to 100]
  Month 36: number analyzed (Participants) | 9
  Month 36 | 100 [66.4 to 100]
  Month 42: number analyzed (Participants) | 5
  Month 42 | 100 [47.8 to 100]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 100 [39.8 to 100]
  Month 54: number analyzed (Participants) | 4
  Month 54 | 100 [39.8 to 100]
  Month 60: number analyzed (Participants) | 3
  Month 60 | 100 [29.2 to 100]
  Month 66: number analyzed (Participants) | 4
  Month 66 | 100 [39.8 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 100 [15.8 to 100]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 100 [2.5 to 100]
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

20. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Pediatric Response (ACR50PR) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: ACR50PR: >=50% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria: physician's global assessment (on 21-circle VAS ranging 0 [no disease activity] to 10 [maximum disease activity],higher score=more severe disease), patient global assessment (on 21-circle VAS ranging 0 [very well] to 10 [very poor],higher score=higher pain), childhood health assessment questionnaire ([CHAQ] Participants >18 years assessed for functional disability, discomfort. Ability to dressing, arising, eat, walk, hygiene, reach, grip, common activities were distributed in 30 items. Each item scored from 0 [no difficulty] to 3 [unable to do]. Highest score for each domain was score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered and ranged from 0 [no difficulty] to 3 [extreme difficulty], where higher scores=more functional disability and discomfort), number of active joints and joints with limited range of motion, C-reactive protein.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 23
  Month 6 | 95.7 [78.1 to 99.9]
  Month 12: number analyzed (Participants) | 60
  Month 12 | 98.3 [91.1 to 100]
  Month 18: number analyzed (Participants) | 61
  Month 18 | 96.7 [88.7 to 99.6]
  Month 24: number analyzed (Participants) | 56
  Month 24 | 98.2 [90.4 to 100]
  Month 30: number analyzed (Participants) | 53
  Month 30 | 98.1 [89.9 to 100]
  Month 36: number analyzed (Participants) | 47
  Month 36 | 100 [92.5 to 100]
  Month 42: number analyzed (Participants) | 46
  Month 42 | 93.5 [82.1 to 98.6]
  Month 48: number analyzed (Participants) | 42
  Month 48 | 97.6 [87.4 to 99.9]
  Month 54: number analyzed (Participants) | 38
  Month 54 | 100 [90.7 to 100]
  Month 60: number analyzed (Participants) | 33
  Month 60 | 100 [89.4 to 100]
  Month 66: number analyzed (Participants) | 31
  Month 66 | 100 [88.8 to 100]
  Month 72: number analyzed (Participants) | 25
  Month 72 | 100 [86.3 to 100]
  Month 78: number analyzed (Participants) | 24
  Month 78 | 100 [85.8 to 100]
  Month 84: number analyzed (Participants) | 21
  Month 84 | 100 [83.9 to 100]
  Month 90: number analyzed (Participants) | 22
  Month 90 | 100 [84.6 to 100]
  Month 96: number analyzed (Participants) | 16
  Month 96 | 100 [79.4 to 100]

21. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Pediatric Response (ACR50PR) at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 20
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 23
  Month 1 | 87.0 [66.4 to 97.2]
  Month 3: number analyzed (Participants) | 15
  Month 3 | 100 [78.2 to 100]
  Month 6: number analyzed (Participants) | 11
  Month 6 | 90.9 [58.7 to 99.8]
  Month 9: number analyzed (Participants) | 9
  Month 9 | 88.9 [51.8 to 99.7]
  Month 12: number analyzed (Participants) | 9
  Month 12 | 88.9 [51.8 to 99.7]
  Month 18: number analyzed (Participants) | 8
  Month 18 | 87.5 [47.3 to 99.7]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 100 [47.8 to 100]
  Month 30: number analyzed (Participants) | 4
  Month 30 | 100 [39.8 to 100]
  Month 36: number analyzed (Participants) | 3
  Month 36 | 100 [29.2 to 100]
  Month 42: number analyzed (Participants) | 4
  Month 42 | 100 [39.8 to 100]
  Month 48: number analyzed (Participants) | 3
  Month 48 | 66.7 [9.4 to 99.2]
  Month 54: number analyzed (Participants) | 1
  Month 54 | 100 [2.5 to 100]
  Month 60: number analyzed (Participants) | 1
  Month 60 | 100 [2.5 to 100]
  Month 66: number analyzed (Participants) | 1
  Month 66 | 100 [2.5 to 100]
  Month 72: number analyzed (Participants) | 1
  Month 72 | 100 [2.5 to 100]
  Month 78: number analyzed (Participants) | 0
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

22. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Pediatric Response (ACR50PR) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Re-treatment Period
Description: ACR50PR:>=50% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria:1)PGA of disease activity(DA),2)PtGA of arthritis pain,3) CHAQ 4)number(no.) of active joints5)no. of joints with limited range of motion 6)C-reactive protein.PGA of DA: 21-circle VAS ranging 0-10, with 0=&10=maximumDA,higher score=more severe disease.PGA:21-circle VAS ranging 0-10,0=very well,10=very poor,higher scores=worsening condition.CHAQ: assessment of functional disability,discomfort. Ability to perform activities:dressing,arising,eating,walking,hygiene,reach,grip, common activities distributed in total of 30 items. Ranging 0=no difficulty;1=some difficulty;2=much difficulty;3=unable to do.Highest score for each domain:score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered.Ranged 0=no difficulty to 3=extreme difficulty;higher scores indicated more functional disability and discomfort. Participants >18 years assessed using CHAQ.
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3: number analyzed (Participants) | 12
  Month 3 | 100 [73.5 to 100]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 100 [73.5 to 100]
  Month 9: number analyzed (Participants) | 12
  Month 9 | 91.7 [61.5 to 99.8]
  Month 12: number analyzed (Participants) | 11
  Month 12 | 90.9 [58.7 to 99.8]
  Month 18: number analyzed (Participants) | 10
  Month 18 | 100 [69.2 to 100]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 87.5 [47.3 to 99.7]
  Month 30: number analyzed (Participants) | 9
  Month 30 | 100 [66.4 to 100]
  Month 36: number analyzed (Participants) | 9
  Month 36 | 100 [66.4 to 100]
  Month 42: number analyzed (Participants) | 5
  Month 42 | 100 [47.8 to 100]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 100 [39.8 to 100]
  Month 54: number analyzed (Participants) | 4
  Month 54 | 100 [39.8 to 100]
  Month 60: number analyzed (Participants) | 3
  Month 60 | 100 [29.2 to 100]
  Month 66: number analyzed (Participants) | 4
  Month 66 | 100 [39.8 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 100 [15.8 to 100]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 100 [2.5 to 100]
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

23. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Pediatric Response (ACR70PR) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: ACR70PR: >=70% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria: physician's global assessment (on 21-circle VAS ranging 0 [no disease activity] to 10 [maximum disease activity],higher score=more severe disease), patient global assessment (on 21-circle VAS ranging 0 [very well] to 10 [very poor],higher score=higher pain), childhood health assessment questionnaire ([CHAQ] Participants >18 years assessed for functional disability, discomfort. Ability to dressing, arising, eat, walk, hygiene, reach, grip, common activities were distributed in 30 items. Each item scored from 0 [no difficulty] to 3 [unable to do]. Highest score for each domain was score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered and ranged from 0 [no difficulty] to 3 [extreme difficulty], where higher scores=more functional disability and discomfort), number of active joints and joints with limited range of motion, C-reactive protein.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 23
  Month 6 | 95.7 [78.1 to 99.9]
  Month 12: number analyzed (Participants) | 62
  Month 12 | 87.1 [76.1 to 94.3]
  Month 18: number analyzed (Participants) | 62
  Month 18 | 88.7 [78.1 to 95.3]
  Month 24: number analyzed (Participants) | 56
  Month 24 | 89.3 [78.1 to 96.0]
  Month 30: number analyzed (Participants) | 52
  Month 30 | 88.5 [76.6 to 95.6]
  Month 36: number analyzed (Participants) | 47
  Month 36 | 89.4 [76.9 to 96.5]
  Month 42: number analyzed (Participants) | 43
  Month 42 | 88.4 [74.9 to 96.1]
  Month 48: number analyzed (Participants) | 41
  Month 48 | 95.1 [83.5 to 99.4]
  Month 54: number analyzed (Participants) | 37
  Month 54 | 100 [90.5 to 100]
  Month 60: number analyzed (Participants) | 33
  Month 60 | 100 [89.4 to 100]
  Month 66: number analyzed (Participants) | 31
  Month 66 | 100 [88.8 to 100]
  Month 72: number analyzed (Participants) | 26
  Month 72 | 96.2 [80.4 to 99.9]
  Month 78: number analyzed (Participants) | 23
  Month 78 | 100 [85.2 to 100]
  Month 84: number analyzed (Participants) | 20
  Month 84 | 100 [83.2 to 100]
  Month 90: number analyzed (Participants) | 22
  Month 90 | 90.9 [70.8 to 98.9]
  Month 96: number analyzed (Participants) | 15
  Month 96 | 93.3 [68.1 to 99.8]

24. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Pediatric Response (ACR70PR) at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 23
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 22
  Month 1 | 77.3 [54.6 to 92.2]
  Month 3: number analyzed (Participants) | 15
  Month 3 | 93.3 [68.1 to 99.8]
  Month 6: number analyzed (Participants) | 11
  Month 6 | 90.9 [58.7 to 99.8]
  Month 9: number analyzed (Participants) | 9
  Month 9 | 88.9 [51.8 to 99.7]
  Month 12: number analyzed (Participants) | 9
  Month 12 | 88.9 [51.8 to 99.7]
  Month 18: number analyzed (Participants) | 7
  Month 18 | 85.7 [42.1 to 99.6]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 100 [47.8 to 100]
  Month 30: number analyzed (Participants) | 4
  Month 30 | 100 [39.8 to 100]
  Month 36: number analyzed (Participants) | 3
  Month 36 | 100 [29.2 to 100]
  Month 42: number analyzed (Participants) | 4
  Month 42 | 100 [39.8 to 100]
  Month 48: number analyzed (Participants) | 3
  Month 48 | 66.7 [9.4 to 99.2]
  Month 54: number analyzed (Participants) | 1
  Month 54 | 100 [2.5 to 100]
  Month 60: number analyzed (Participants) | 1
  Month 60 | 100 [2.5 to 100]
  Month 66: number analyzed (Participants) | 1
  Month 66 | 100 [2.5 to 100]
  Month 72: number analyzed (Participants) | 1
  Month 72 | 100 [2.5 to 100]
  Month 78: number analyzed (Participants) | 0
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

25. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Pediatric Response (ACR70PR) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 23
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3: number analyzed (Participants) | 12
  Month 3 | 91.7 [61.5 to 99.8]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 83.3 [51.6 to 97.9]
  Month 9: number analyzed (Participants) | 11
  Month 9 | 81.8 [48.2 to 97.7]
  Month 12: number analyzed (Participants) | 11
  Month 12 | 81.8 [48.2 to 97.7]
  Month 18: number analyzed (Participants) | 10
  Month 18 | 80.0 [44.4 to 97.5]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 75.0 [34.9 to 96.8]
  Month 30: number analyzed (Participants) | 9
  Month 30 | 66.7 [29.9 to 92.5]
  Month 36: number analyzed (Participants) | 9
  Month 36 | 88.9 [51.8 to 99.7]
  Month 42: number analyzed (Participants) | 6
  Month 42 | 83.3 [35.9 to 99.6]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 100 [39.8 to 100]
  Month 54: number analyzed (Participants) | 4
  Month 54 | 100 [39.8 to 100]
  Month 60: number analyzed (Participants) | 3
  Month 60 | 100 [29.2 to 100]
  Month 66: number analyzed (Participants) | 3
  Month 66 | 100 [29.2 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 100 [15.8 to 100]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 100 [2.5 to 100]
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

26. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 90% (ACR90) Pediatric Response (ACR90PR) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: ACR90PR: >=90% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria: physician's global assessment (on 21-circle VAS ranging 0 [no disease activity] to 10 [maximum disease activity],higher score=more severe disease), patient global assessment (on 21-circle VAS ranging 0 [very well] to 10 [very poor],higher score=higher pain), childhood health assessment questionnaire ([CHAQ] Participants >18 years assessed for functional disability, discomfort. Ability to dressing, arising, eat, walk, hygiene, reach, grip, common activities were distributed in 30 items. Each item scored from 0 [no difficulty] to 3 [unable to do]. Highest score for each domain was score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered and ranged from 0 [no difficulty] to 3 [extreme difficulty], where higher scores=more functional disability and discomfort), number of active joints and joints with limited range of motion, C-reactive protein.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 25
  Month 6 | 64.0 [42.5 to 82.0]
  Month 12: number analyzed (Participants) | 57
  Month 12 | 70.2 [56.6 to 81.6]
  Month 18: number analyzed (Participants) | 62
  Month 18 | 72.6 [59.8 to 83.1]
  Month 24: number analyzed (Participants) | 54
  Month 24 | 64.8 [50.6 to 77.3]
  Month 30: number analyzed (Participants) | 52
  Month 30 | 63.5 [49.0 to 76.4]
  Month 36: number analyzed (Participants) | 45
  Month 36 | 71.1 [55.7 to 83.6]
  Month 42: number analyzed (Participants) | 43
  Month 42 | 67.4 [51.5 to 80.9]
  Month 48: number analyzed (Participants) | 41
  Month 48 | 65.9 [49.4 to 79.9]
  Month 54: number analyzed (Participants) | 31
  Month 54 | 77.4 [58.9 to 90.4]
  Month 60: number analyzed (Participants) | 29
  Month 60 | 89.7 [72.6 to 97.8]
  Month 66: number analyzed (Participants) | 24
  Month 66 | 87.5 [67.6 to 97.3]
  Month 72: number analyzed (Participants) | 24
  Month 72 | 75.0 [53.3 to 90.2]
  Month 78: number analyzed (Participants) | 17
  Month 78 | 100 [80.5 to 100]
  Month 84: number analyzed (Participants) | 18
  Month 84 | 77.8 [52.4 to 93.6]
  Month 90: number analyzed (Participants) | 20
  Month 90 | 90.0 [68.3 to 98.8]
  Month 96: number analyzed (Participants) | 15
  Month 96 | 86.7 [59.5 to 98.3]

27. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 90% (ACR90) Pediatric Response (ACR90PR) at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 26
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 21
  Month 1 | 66.7 [43.0 to 85.4]
  Month 3: number analyzed (Participants) | 14
  Month 3 | 71.4 [41.9 to 91.6]
  Month 6: number analyzed (Participants) | 10
  Month 6 | 70.0 [34.8 to 93.3]
  Month 9: number analyzed (Participants) | 8
  Month 9 | 75.0 [34.9 to 96.8]
  Month 12: number analyzed (Participants) | 8
  Month 12 | 87.5 [47.3 to 99.7]
  Month 18: number analyzed (Participants) | 8
  Month 18 | 75.0 [34.9 to 96.8]
  Month 24: number analyzed (Participants) | 4
  Month 24 | 100 [39.8 to 100]
  Month 30: number analyzed (Participants) | 4
  Month 30 | 100 [39.8 to 100]
  Month 36: number analyzed (Participants) | 4
  Month 36 | 75.0 [19.4 to 99.4]
  Month 42: number analyzed (Participants) | 4
  Month 42 | 75.0 [19.4 to 99.4]
  Month 48: number analyzed (Participants) | 3
  Month 48 | 66.7 [9.4 to 99.2]
  Month 54: number analyzed (Participants) | 2
  Month 54 | 50.0 [1.3 to 98.7]
  Month 60: number analyzed (Participants) | 1
  Month 60 | 100 [2.5 to 100]
  Month 66: number analyzed (Participants) | 1
  Month 66 | 100 [2.5 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 50.0 [1.3 to 98.7]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 0.0 [0.0 to 97.5]
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

28. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 90% (ACR90) Pediatric Response (ACR90PR) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 26
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3: number analyzed (Participants) | 11
  Month 3 | 63.6 [30.8 to 89.1]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 66.7 [34.9 to 90.1]
  Month 9: number analyzed (Participants) | 12
  Month 9 | 66.7 [34.9 to 90.1]
  Month 12: number analyzed (Participants) | 10
  Month 12 | 70.0 [34.8 to 93.3]
  Month 18: number analyzed (Participants) | 8
  Month 18 | 75.0 [34.9 to 96.8]
  Month 24: number analyzed (Participants) | 7
  Month 24 | 57.1 [18.4 to 90.1]
  Month 30: number analyzed (Participants) | 8
  Month 30 | 62.5 [24.5 to 91.5]
  Month 36: number analyzed (Participants) | 8
  Month 36 | 87.5 [47.3 to 99.7]
  Month 42: number analyzed (Participants) | 5
  Month 42 | 60.0 [14.7 to 94.7]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 25.0 [0.6 to 80.6]
  Month 54: number analyzed (Participants) | 4
  Month 54 | 50.0 [6.8 to 93.2]
  Month 60: number analyzed (Participants) | 4
  Month 60 | 50.0 [6.8 to 93.2]
  Month 66: number analyzed (Participants) | 4
  Month 66 | 50.0 [6.8 to 93.2]
  Month 72: number analyzed (Participants) | 3
  Month 72 | 33.3 [0.8 to 90.6]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 100 [2.5 to 100]
  Month 84: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

29. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 100% (ACR100) Pediatric Response (ACR100PR) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: ACR100PR: 100% improvement from baseline in 3 of 6 criteria with worsening >30% in no more than 1 of 6 criteria: physician's global assessment (on 21-circle VAS ranging 0 [no disease activity] to 10 [maximum disease activity],higher score=more severe disease), patient global assessment (on 21-circle VAS ranging 0 [very well] to 10 [very poor],higher score=higher pain), childhood health assessment questionnaire ([CHAQ] Participants >18 years assessed for functional disability, discomfort. Ability to dressing, arising, eat, walk, hygiene, reach, grip, common activities were distributed in 30 items. Each item scored from 0 [no difficulty] to 3 [unable to do]. Highest score for each domain was score for that domain. Overall CHAQ score=sum of domain scores/number of domains answered and ranged from 0 [no difficulty] to 3 [extreme difficulty], where higher scores=more functional disability and discomfort), number of active joints and joints with limited range of motion, C-reactive protein.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 25
  Month 6 | 44.0 [24.4 to 65.1]
  Month 12: number analyzed (Participants) | 54
  Month 12 | 51.9 [37.8 to 65.7]
  Month 18: number analyzed (Participants) | 60
  Month 18 | 55.0 [41.6 to 67.9]
  Month 24: number analyzed (Participants) | 55
  Month 24 | 45.5 [32.0 to 59.4]
  Month 30: number analyzed (Participants) | 52
  Month 30 | 40.4 [27.0 to 54.9]
  Month 36: number analyzed (Participants) | 36
  Month 36 | 52.8 [35.5 to 69.6]
  Month 42: number analyzed (Participants) | 37
  Month 42 | 48.6 [31.9 to 65.6]
  Month 48: number analyzed (Participants) | 35
  Month 48 | 48.6 [31.4 to 66.0]
  Month 54: number analyzed (Participants) | 30
  Month 54 | 56.7 [37.4 to 74.5]
  Month 60: number analyzed (Participants) | 24
  Month 60 | 62.5 [40.6 to 81.2]
  Month 66: number analyzed (Participants) | 21
  Month 66 | 57.1 [34.0 to 78.2]
  Month 72: number analyzed (Participants) | 18
  Month 72 | 38.9 [17.3 to 64.3]
  Month 78: number analyzed (Participants) | 16
  Month 78 | 75.0 [47.6 to 92.7]
  Month 84: number analyzed (Participants) | 15
  Month 84 | 53.3 [26.6 to 78.7]
  Month 90: number analyzed (Participants) | 14
  Month 90 | 71.4 [41.9 to 91.6]
  Month 96: number analyzed (Participants) | 9
  Month 96 | 77.8 [40.0 to 97.2]

30. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 100% (ACR100) Pediatric Response (ACR100PR) at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 29
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 21
  Month 1 | 61.9 [38.4 to 81.9]
  Month 3: number analyzed (Participants) | 14
  Month 3 | 64.3 [35.1 to 87.2]
  Month 6: number analyzed (Participants) | 11
  Month 6 | 63.6 [30.8 to 89.1]
  Month 9: number analyzed (Participants) | 9
  Month 9 | 66.7 [29.9 to 92.5]
  Month 12: number analyzed (Participants) | 9
  Month 12 | 77.8 [40.0 to 97.2]
  Month 18: number analyzed (Participants) | 9
  Month 18 | 66.7 [29.9 to 92.5]
  Month 24: number analyzed (Participants) | 5
  Month 24 | 80.0 [28.4 to 99.5]
  Month 30: number analyzed (Participants) | 5
  Month 30 | 80.0 [28.4 to 99.5]
  Month 36: number analyzed (Participants) | 4
  Month 36 | 75.0 [19.4 to 99.4]
  Month 42: number analyzed (Participants) | 5
  Month 42 | 60.0 [14.7 to 94.7]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 50.0 [6.8 to 93.2]
  Month 54: number analyzed (Participants) | 2
  Month 54 | 50.0 [1.3 to 98.7]
  Month 60: number analyzed (Participants) | 1
  Month 60 | 100 [2.5 to 100]
  Month 66: number analyzed (Participants) | 1
  Month 66 | 100 [2.5 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 50.0 [1.3 to 98.7]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 0.0 [0.0 to 97.5]
  Month 84: number analyzed (Participants) | 0
  Month 90: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

31. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 100% (ACR100) Pediatric Response (ACR100PR) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 29
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3: number analyzed (Participants) | 11
  Month 3 | 54.5 [23.4 to 83.3]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 50.0 [21.1 to 78.9]
  Month 9: number analyzed (Participants) | 11
  Month 9 | 63.6 [30.8 to 89.1]
  Month 12: number analyzed (Participants) | 8
  Month 12 | 62.5 [24.5 to 91.5]
  Month 18: number analyzed (Participants) | 8
  Month 18 | 75.0 [34.9 to 96.8]
  Month 24: number analyzed (Participants) | 7
  Month 24 | 57.1 [18.4 to 90.1]
  Month 30: number analyzed (Participants) | 7
  Month 30 | 57.1 [18.4 to 90.1]
  Month 36: number analyzed (Participants) | 8
  Month 36 | 87.5 [47.3 to 99.7]
  Month 42: number analyzed (Participants) | 5
  Month 42 | 60.0 [14.7 to 94.7]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 25.0 [0.6 to 80.6]
  Month 54: number analyzed (Participants) | 4
  Month 54 | 50.0 [6.8 to 93.2]
  Month 60: number analyzed (Participants) | 4
  Month 60 | 50.0 [6.8 to 93.2]
  Month 66: number analyzed (Participants) | 4
  Month 66 | 50.0 [6.8 to 93.2]
  Month 72: number analyzed (Participants) | 3
  Month 72 | 33.3 [0.8 to 90.6]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 100 [2.5 to 100]
  Month 84: number analyzed (Participants) | 0
  Month 90: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

32. Secondary Outcome: Change From Baseline (of Parent Study) in Physician's Global Assessment of Disease Activity Score at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96 of Extension Study: Active Treatment Period
Description: PGA of disease activity was measured on a 21-circle Visual Analog Scale (VAS) ranging from 0 to 10, with 0 = no disease activity and 10= maximum disease activity, where higher score indicated more severe disease.
Time Frame: Baseline of the parent study; Month 12, 24, 36, 48, 60, 72, 84 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 96
  Change at Month 6 of extension study | -4.51 (1.63)
  Change at Month 12 of extension study: number analyzed (Participants) | 86
  Change at Month 12 of extension study | -4.66 (1.83)
  Change at Month 18 of extension study: number analyzed (Participants) | 73
  Change at Month 18 of extension study | -4.71 (2.10)
  Change at Month 24 of extension study: number analyzed (Participants) | 63
  Change at Month 24 of extension study | -4.67 (1.73)
  Change at Month 30 of extension study: number analyzed (Participants) | 60
  Change at Month 30 of extension study | -4.69 (1.94)
  Change at Month 36 of extension study: number analyzed (Participants) | 57
  Change at Month 36 of extension study | -4.75 (1.72)
  Change at Month 42 of extension study: number analyzed (Participants) | 53
  Change at Month 42 of extension study | -4.71 (2.00)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -4.80 (1.79)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -5.05 (1.82)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -5.19 (1.64)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -5.10 (1.80)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -5.21 (1.81)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -5.15 (1.58)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -5.17 (1.69)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -5.15 (1.67)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -5.11 (1.65)

33. Secondary Outcome: Change From Baseline (of Parent Study) in Physician's Global Assessment of Disease Activity Score at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: PGA of disease activity was measured on a 21-circle VAS ranging from 0 to 10, with 0 = no disease activity and 10= maximum disease activity, where higher score indicated more severe disease.
Time Frame: Baseline of the parent study; Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1 of extension study: number analyzed (Participants) | 24
  Change at Month 1 of extension study | -4.92 (2.35)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -4.70 (2.40)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -5.50 (1.99)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -5.09 (2.17)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -5.30 (2.14)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -5.15 (2.42)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -4.88 (2.05)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -4.50 (1.89)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -4.50 (1.89)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -4.33 (2.09)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -5.13 (2.10)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -5.33 (2.52)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -5.67 (2.08)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -6.00 (2.83)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -4.50 (2.12)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -2.50
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

34. Secondary Outcome: Change From Baseline (of Parent Study) in Physician's Global Assessment of Disease Activity Score at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 33
Time Frame: Baseline of the parent study; Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3 of extension study | -3.73 (1.51)
  Change at Month 6 of extension study | -4.19 (1.53)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -4.13 (2.05)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -3.82 (2.69)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -3.85 (2.17)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -3.81 (2.55)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -3.94 (2.30)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -4.11 (2.16)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -4.14 (2.53)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -3.58 (1.86)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -3.42 (1.43)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -2.60 (0.74)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -2.63 (0.85)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -2.33 (0.76)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -3.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

35. Secondary Outcome: Change From Baseline (of Parent Study) in Patient/Parent Global Assessment Score at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: Patient/Parent Global Assessment was assessed by the participant's parent using a 21-circle VAS ranging from 0 to 10, with 0 = very well and 10 = very poor, where higher scores indicated worsening of condition.
Time Frame: Baseline of the parent study; Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 96
  Change at Month 6 of extension study | -3.93 (2.31)
  Change at Month 12 of extension study: number analyzed (Participants) | 85
  Change at Month 12 of extension study | -3.79 (2.49)
  Change at Month 18 of extension study: number analyzed (Participants) | 71
  Change at Month 18 of extension study | -4.13 (2.49)
  Change at Month 24 of extension study: number analyzed (Participants) | 64
  Change at Month 24 of extension study | -4.18 (2.60)
  Change at Month 30 of extension study: number analyzed (Participants) | 61
  Change at Month 30 of extension study | -4.38 (2.27)
  Change at Month 36 of extension study: number analyzed (Participants) | 57
  Change at Month 36 of extension study | -4.20 (2.24)
  Change at Month 42 of extension study: number analyzed (Participants) | 51
  Change at Month 42 of extension study | -4.05 (2.85)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -4.37 (2.29)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -4.74 (2.33)
  Change at Month 60 of extension study: number analyzed (Participants) | 38
  Change at Month 60 of extension study | -4.45 (2.57)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -4.54 (2.54)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -4.50 (2.63)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -4.62 (1.87)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -4.57 (1.90)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -4.72 (2.08)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -4.85 (2.11)

36. Secondary Outcome: Change From Baseline (of Parent Study) in Patient/Parent Global Assessment Score at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 35
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1 of extension study: number analyzed (Participants) | 24
  Change at Month 1 of extension study | -4.38 (2.77)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -3.97 (2.88)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -5.04 (2.58)
  Change at Month 9 of extension study: number analyzed (Participants) | 10
  Change at Month 9 of extension study | -4.65 (2.73)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -4.60 (2.77)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -4.50 (2.84)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -4.63 (2.75)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -4.07 (2.41)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -4.14 (2.66)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -3.83 (2.77)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -3.25 (3.77)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -4.00 (3.77)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -4.00 (4.00)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -4.00 (5.66)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -4.25 (5.30)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -0.50
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

37. Secondary Outcome: Change From Baseline (of Parent Study) in Patient/Parent Global Assessment Score at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 35
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3 of extension study | -2.81 (1.95)
  Change at Month 6 of extension study | -2.73 (2.26)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -2.83 (2.79)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -2.86 (3.03)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -2.65 (2.65)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -2.81 (2.90)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -2.44 (2.86)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -2.83 (2.63)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -2.93 (3.06)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -2.17 (2.36)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -2.33 (1.99)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -1.30 (1.20)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -1.13 (0.95)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -1.50 (1.00)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -2.50
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

38. Secondary Outcome: Change From Baseline (of Parent Study) in Childhood Health Assessment Questionnaire (CHAQ) Score for Participants at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: CHAQ: parent-administered, valid assessment of functional disability, discomfort in pediatrics with rheumatic diseases. Parents report participant's ability to perform activities in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, common activities distributed in total of 30 items. Each item is scored on 4-point Likert scale: 0=no difficulty;1=some difficulty;2=much difficulty;3=unable to do. Highest score reported for each domain is score for that domain. Overall CHAQ score was calculated as sum of domain scores divided by number of domains answered and ranged from 0=no difficulty to 3=extreme difficulty, where higher scores indicated more functional disability and discomfort in pediatrics with rheumatic disease. Participants below 18 years of age were assessed using CHAQ.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 74
  Change at Month 6 of extension study | -0.66 (0.60)
  Change at Month 12 of extension study: number analyzed (Participants) | 62
  Change at Month 12 of extension study | -0.71 (0.58)
  Change at Month 18 of extension study: number analyzed (Participants) | 46
  Change at Month 18 of extension study | -0.72 (0.56)
  Change at Month 24 of extension study: number analyzed (Participants) | 37
  Change at Month 24 of extension study | -0.81 (0.59)
  Change at Month 30 of extension study: number analyzed (Participants) | 32
  Change at Month 30 of extension study | -0.82 (0.57)
  Change at Month 36 of extension study: number analyzed (Participants) | 22
  Change at Month 36 of extension study | -0.86 (0.60)
  Change at Month 42 of extension study: number analyzed (Participants) | 21
  Change at Month 42 of extension study | -0.81 (0.67)
  Change at Month 48 of extension study: number analyzed (Participants) | 16
  Change at Month 48 of extension study | -0.97 (0.69)
  Change at Month 54 of extension study: number analyzed (Participants) | 10
  Change at Month 54 of extension study | -1.15 (0.75)
  Change at Month 60 of extension study: number analyzed (Participants) | 8
  Change at Month 60 of extension study | -1.33 (0.81)
  Change at Month 66 of extension study: number analyzed (Participants) | 7
  Change at Month 66 of extension study | -1.48 (0.75)
  Change at Month 72 of extension study: number analyzed (Participants) | 6
  Change at Month 72 of extension study | -1.50 (0.76)
  Change at Month 78 of extension study: number analyzed (Participants) | 5
  Change at Month 78 of extension study | -1.40 (0.71)
  Change at Month 84 of extension study: number analyzed (Participants) | 4
  Change at Month 84 of extension study | -1.41 (0.83)
  Change at Month 90 of extension study: number analyzed (Participants) | 4
  Change at Month 90 of extension study | -1.41 (0.83)
  Change at Month 96 of extension study: number analyzed (Participants) | 2
  Change at Month 96 of extension study | -1.13 (1.24)

39. Secondary Outcome: Change From Baseline (of Parent Study) in Childhood Health Assessment Questionnaire (CHAQ) Score for Participants at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 38
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1 of extension study: number analyzed (Participants) | 15
  Change at Month 1 of extension study | -0.81 (0.86)
  Change at Month 3 of extension study: number analyzed (Participants) | 9
  Change at Month 3 of extension study | -0.90 (0.82)
  Change at Month 6 of extension study: number analyzed (Participants) | 6
  Change at Month 6 of extension study | -1.04 (0.95)
  Change at Month 9 of extension study: number analyzed (Participants) | 6
  Change at Month 9 of extension study | -1.04 (1.09)
  Change at Month 12 of extension study: number analyzed (Participants) | 15
  Change at Month 12 of extension study | -1.15 (1.16)
  Change at Month 18 of extension study: number analyzed (Participants) | 5
  Change at Month 18 of extension study | -1.15 (1.16)
  Change at Month 24 of extension study: number analyzed (Participants) | 1
  Change at Month 24 of extension study | -2.13
  Change at Month 30 of extension study: number analyzed (Participants) | 1
  Change at Month 30 of extension study | -2.13
  Change at Month 36 of extension study: number analyzed (Participants) | 1
  Change at Month 36 of extension study | -2.13
  Change at Month 42 of extension study: number analyzed (Participants) | 1
  Change at Month 42 of extension study | -2.13
  Change at Month 48 of extension study: number analyzed (Participants) | 1
  Change at Month 48 of extension study | -2.13
  Change at Month 54 of extension study: number analyzed (Participants) | 1
  Change at Month 54 of extension study | -2.13
  Change at Month 60 of extension study: number analyzed (Participants) | 1
  Change at Month 60 of extension study | -2.13
  Change at Month 66 of extension study: number analyzed (Participants) | 1
  Change at Month 66 of extension study | -2.13
  Change at Month 72 of extension study: number analyzed (Participants) | 1
  Change at Month 72 of extension study | -2.13
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -2.13
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

40. Secondary Outcome: Change From Baseline (of Parent Study) in Childhood Health Assessment Questionnaire (CHAQ) Score for Participants at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 38
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3 of extension study: number analyzed (Participants) | 11
  Change at Month 3 of extension study | -0.65 (0.66)
  Change at Month 6 of extension study: number analyzed (Participants) | 10
  Change at Month 6 of extension study | -0.66 (0.73)
  Change at Month 9 of extension study: number analyzed (Participants) | 8
  Change at Month 9 of extension study | -0.78 (0.79)
  Change at Month 12 of extension study: number analyzed (Participants) | 8
  Change at Month 12 of extension study | -0.80 (0.78)
  Change at Month 18 of extension study: number analyzed (Participants) | 8
  Change at Month 18 of extension study | -0.78 (0.79)
  Change at Month 24 of extension study: number analyzed (Participants) | 7
  Change at Month 24 of extension study | -0.75 (0.85)
  Change at Month 30 of extension study: number analyzed (Participants) | 6
  Change at Month 30 of extension study | -0.79 (0.92)
  Change at Month 36 of extension study: number analyzed (Participants) | 6
  Change at Month 36 of extension study | -0.88 (0.87)
  Change at Month 42 of extension study: number analyzed (Participants) | 4
  Change at Month 42 of extension study | -0.94 (1.11)
  Change at Month 48 of extension study: number analyzed (Participants) | 3
  Change at Month 48 of extension study | -0.42 (0.62)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -0.42 (0.62)
  Change at Month 60 of extension study: number analyzed (Participants) | 2
  Change at Month 60 of extension study | -0.06 (0.09)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -0.06 (0.09)
  Change at Month 72 of extension study: number analyzed (Participants) | 1
  Change at Month 72 of extension study | -0.13
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

41. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score for Participants Years at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: HAQ is a self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ total score range from 0 to 3, where 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; > 1=significant functional limitation. Participants aged 18 years or above were assessed using HAQ scores.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6: number analyzed (Participants) | 10
  Change at Month 6 | 0.09 (0.19)
  Change at Month 12: number analyzed (Participants) | 10
  Change at Month 12 | 0.10 (0.16)
  Change at Month 18: number analyzed (Participants) | 8
  Change at Month 18 | 0.09 (0.19)
  Change at Month 24: number analyzed (Participants) | 6
  Change at Month 24 | 0.13 (0.19)
  Change at Month 30: number analyzed (Participants) | 6
  Change at Month 30 | 0.15 (0.23)
  Change at Month 36: number analyzed (Participants) | 6
  Change at Month 36 | 0.17 (0.27)
  Change at Month 42: number analyzed (Participants) | 6
  Change at Month 42 | 0.13 (0.25)
  Change at Month 48: number analyzed (Participants) | 6
  Change at Month 48 | 0.17 (0.27)
  Change at Month 54: number analyzed (Participants) | 5
  Change at Month 54 | 0.13 (0.18)
  Change at Month 60: number analyzed (Participants) | 5
  Change at Month 60 | 0.18 (0.24)
  Change at Month 66: number analyzed (Participants) | 3
  Change at Month 66 | 0.33 (0.31)
  Change at Month 72: number analyzed (Participants) | 3
  Change at Month 72 | 0.29 (0.26)
  Change at Month 78: number analyzed (Participants) | 3
  Change at Month 78 | 0.13 (0.22)
  Change at Month 84: number analyzed (Participants) | 3
  Change at Month 84 | 0.25 (0.33)
  Change at Month 90: number analyzed (Participants) | 2
  Change at Month 90 | 0.13 (0.18)
  Change at Month 96: number analyzed (Participants) | 1
  Change at Month 96 | 0.63

42. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score for Participants at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 41
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1: number analyzed (Participants) | 9
  Change at Month 1 | 0.00 (0.00)
  Change at Month 3: number analyzed (Participants) | 6
  Change at Month 3 | 0.02 (0.05)
  Change at Month 6: number analyzed (Participants) | 5
  Change at Month 6 | 0.03 (0.06)
  Change at Month 9: number analyzed (Participants) | 4
  Change at Month 9 | 0.00 (0.00)
  Change at Month 12: number analyzed (Participants) | 4
  Change at Month 12 | 0.00 (0.00)
  Change at Month 18: number analyzed (Participants) | 4
  Change at Month 18 | 0.00 (0.00)
  Change at Month 24: number analyzed (Participants) | 4
  Change at Month 24 | 0.00 (0.00)
  Change at Month 30: number analyzed (Participants) | 3
  Change at Month 30 | 0.04 (0.07)
  Change at Month 36: number analyzed (Participants) | 3
  Change at Month 36 | 0.00 (0.00)
  Change at Month 42: number analyzed (Participants) | 3
  Change at Month 42 | 0.00 (0.00)
  Change at Month 48: number analyzed (Participants) | 1
  Change at Month 48 | 0.00 (0.00)
  Change at Month 54: number analyzed (Participants) | 1
  Change at Month 54 | 0.00 (0.00)
  Change at Month 60: number analyzed (Participants) | 1
  Change at Month 60 | 0.00 (0.00)
  Change at Month 66: number analyzed (Participants) | 0
  Change at Month 72: number analyzed (Participants) | 0
  Change at Month 78: number analyzed (Participants) | 0
  Change at Month 84: number analyzed (Participants) | 0
  Change at Month 90: number analyzed (Participants) | 0
  Change at Month 96: number analyzed (Participants) | 0

43. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score for Participants at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 41
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3: number analyzed (Participants) | 2
  Change at Month 3 | -0.81 (0.09)
  Change at Month 6: number analyzed (Participants) | 2
  Change at Month 6 | -0.81 (0.09)
  Change at Month 9: number analyzed (Participants) | 3
  Change at Month 9 | -0.42 (0.69)
  Change at Month 12: number analyzed (Participants) | 2
  Change at Month 12 | -0.81 (0.09)
  Change at Month 18: number analyzed (Participants) | 1
  Change at Month 18 | -0.75
  Change at Month 24: number analyzed (Participants) | 1
  Change at Month 24 | -0.75
  Change at Month 30: number analyzed (Participants) | 1
  Change at Month 30 | -0.75
  Change at Month 36: number analyzed (Participants) | 1
  Change at Month 36 | -0.75
  Change at Month 42: number analyzed (Participants) | 1
  Change at Month 42 | -0.75
  Change at Month 48: number analyzed (Participants) | 1
  Change at Month 48 | -0.75
  Change at Month 54: number analyzed (Participants) | 1
  Change at Month 54 | -0.75
  Change at Month 60: number analyzed (Participants) | 1
  Change at Month 60 | -0.75
  Change at Month 66: number analyzed (Participants) | 1
  Change at Month 66 | -0.75
  Change at Month 72: number analyzed (Participants) | 1
  Change at Month 72 | -0.75
  Change at Month 78: number analyzed (Participants) | 1
  Change at Month 78 | -0.75
  Change at Month 84: number analyzed (Participants) | 0
  Change at Month 90: number analyzed (Participants) | 0
  Change at Month 96: number analyzed (Participants) | 0

44. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Active Arthritis at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: Joints with active arthritis were defined as joints that were swollen or, in the absence of swelling, joints with limited range of motion accompanied by pain and/or tenderness.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Joints
  Change at Month 6 of extension study: number analyzed (Participants) | 25
  Change at Month 6 of extension study | -7.00 (5.92)
  Change at Month 12 of extension study: number analyzed (Participants) | 67
  Change at Month 12 of extension study | -6.94 (5.59)
  Change at Month 18 of extension study: number analyzed (Participants) | 72
  Change at Month 18 of extension study | -6.82 (5.39)
  Change at Month 24 of extension study: number analyzed (Participants) | 65
  Change at Month 24 of extension study | -6.48 (4.64)
  Change at Month 30 of extension study: number analyzed (Participants) | 61
  Change at Month 30 of extension study | -6.43 (4.41)
  Change at Month 36 of extension study: number analyzed (Participants) | 56
  Change at Month 36 of extension study | -6.82 (4.46)
  Change at Month 42 of extension study: number analyzed (Participants) | 52
  Change at Month 42 of extension study | -6.98 (4.78)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -7.27 (4.56)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -7.71 (4.93)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -7.74 (4.51)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -7.56 (4.35)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -7.56 (4.24)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -7.40 (3.83)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -7.14 (3.74)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -7.37 (3.69)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -7.17 (3.58)

45. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Active Arthritis at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 44
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Joints
  Change at Month 1 of extension study: number analyzed (Participants) | 24
  Change at Month 1 of extension study | -6.96 (5.38)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -8.53 (5.48)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -8.50 (4.80)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -8.73 (4.96)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -8.70 (5.27)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -8.40 (5.19)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -8.38 (4.69)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -7.00 (2.83)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -6.86 (3.02)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -7.17 (2.99)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -6.75 (2.75)
  Change at Month 53 of extension study: number analyzed (Participants) | 3
  Change at Month 53 of extension study | -6.67 (3.06)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -7.00 (3.00)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -8.50 (2.12)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -7.50 (2.12)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -5.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

46. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Active Arthritis at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 44
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Joints
  Change at Month 3 of extension study | -6.31 (4.31)
  Change at Month 6 of extension study | -6.46 (4.29)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -6.17 (4.73)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -6.18 (4.92)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -6.60 (4.97)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -5.63 (2.62)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -5.33 (2.50)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -5.67 (2.35)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -5.86 (2.54)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -5.33 (1.97)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -5.33 (1.97)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -4.60 (0.89)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -4.75 (0.96)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -4.33 (0.58)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -5.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

47. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Limited Motion at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: Total number of joints with limited range of motion was the number of joints with limited range of motion. It was defined as 69*(total number of joints with score of limited range of motion greater than zero)/number of non-missing limited range of motions. Joint replacement (JR) and not evaluable (NE) were treated as missing. If more than 34 scores of limited range of motion were missing, then the total number of joints with limited range of motion was defined as missing.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Joints
  Change at Month 6 of extension study: number analyzed (Participants) | 25
  Change at Month 6 of extension study | -4.80 (5.39)
  Change at Month 12 of extension study: number analyzed (Participants) | 67
  Change at Month 12 of extension study | -5.51 (5.18)
  Change at Month 18 of extension study: number analyzed (Participants) | 72
  Change at Month 18 of extension study | -5.32 (5.27)
  Change at Month 24 of extension study: number analyzed (Participants) | 65
  Change at Month 24 of extension study | -5.12 (4.83)
  Change at Month 30 of extension study: number analyzed (Participants) | 61
  Change at Month 30 of extension study | -5.03 (4.19)
  Change at Month 36 of extension study: number analyzed (Participants) | 56
  Change at Month 36 of extension study | -5.23 (4.26)
  Change at Month 42 of extension study: number analyzed (Participants) | 52
  Change at Month 42 of extension study | -5.63 (4.69)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -5.90 (4.33)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -6.57 (4.71)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -6.38 (4.02)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -6.64 (3.86)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -6.71 (4.11)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -6.90 (4.15)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -6.45 (4.15)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -6.63 (3.82)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -6.57 (3.72)

48. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Limited Motion at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: Total number of joints with limited range of motion was the number of joints with limited range of motion. It was defined as 69*(total number of joints with score of limited range of motion greater than zero)/number of non-missing limited range of motions. JR and NE were treated as missing. If more than 34 scores of limited range of motion were missing, then the total number of joints with limited range of motion was defined as missing.
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Joints
  Change at Month 1 of extension study: number analyzed (Participants) | 24
  Change at Month 1 of extension study | -5.38 (4.68)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -5.60 (5.15)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -5.67 (3.68)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -5.36 (3.70)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -5.40 (4.01)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -5.10 (3.54)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -4.75 (3.20)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -4.71 (3.45)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -4.71 (3.45)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -4.83 (3.76)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -3.25 (4.03)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -2.00 (1.00)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -1.67 (1.15)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -2.00 (1.41)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -2.00 (1.41)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | 1.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

49. Secondary Outcome: Change From Baseline (of Parent Study) in Number of Joints With Limited Motion at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 48
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Joints
  Change at Month 3 of extension study | -5.15 (4.83)
  Change at Month 6 of extension study | -5.46 (4.82)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -4.75 (5.59)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -5.45 (5.48)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -5.60 (5.60)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -3.88 (4.45)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -3.78 (4.18)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -4.44 (3.97)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -4.71 (4.39)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -3.83 (3.87)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -3.83 (3.87)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -2.80 (2.86)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -3.00 (2.94)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -2.00 (2.65)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -1.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

50. Secondary Outcome: Change From Baseline (of Parent Study) in C-reactive Protein at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milligram/Liter
Arm/Group | Etanercept
Number analyzed (Participants) | 99
milligram/Liter
  Change at Month 6 of extension study: number analyzed (Participants) | 93
  Change at Month 6 of extension study | -3.71 (12.20)
  Change at Month 12 of extension study: number analyzed (Participants) | 82
  Change at Month 12 of extension study | -3.37 (13.01)
  Change at Month 18 of extension study: number analyzed (Participants) | 71
  Change at Month 18 of extension study | -3.82 (15.17)
  Change at Month 24 of extension study: number analyzed (Participants) | 64
  Change at Month 24 of extension study | -4.00 (13.89)
  Change at Month 30 of extension study: number analyzed (Participants) | 61
  Change at Month 30 of extension study | -3.89 (12.93)
  Change at Month 36 of extension study: number analyzed (Participants) | 55
  Change at Month 36 of extension study | -3.52 (14.91)
  Change at Month 42 of extension study: number analyzed (Participants) | 53
  Change at Month 42 of extension study | -1.96 (22.18)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -5.01 (14.61)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -5.79 (15.49)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -3.25 (13.28)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -4.39 (13.61)
  Change at Month 72 of extension study: number analyzed (Participants) | 31
  Change at Month 72 of extension study | -4.64 (13.76)
  Change at Month 78 of extension study: number analyzed (Participants) | 27
  Change at Month 78 of extension study | -4.31 (11.17)
  Change at Month 84 of extension study: number analyzed (Participants) | 28
  Change at Month 84 of extension study | -4.52 (15.32)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -5.37 (15.17)
  Change at Month 96 of extension study: number analyzed (Participants) | 22
  Change at Month 96 of extension study | -0.59 (22.63)

51. Secondary Outcome: Change From Baseline (of Parent Study) in C-reactive Protein at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 50
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milligram/Liter
Arm/Group | Etanercept
Number analyzed (Participants) | 30
milligram/Liter
  Change at Month 1 of extension study: number analyzed (Participants) | 22
  Change at Month 1 of extension study | -0.99 (14.06)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -2.47 (6.73)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -3.01 (6.89)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -0.27 (1.26)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -0.25 (1.19)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | 0.07 (2.07)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | 0.14 (1.61)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | 1.19 (2.48)
  Change at Month 36 of extension study: number analyzed (Participants) | 6
  Change at Month 36 of extension study | 0.15 (1.13)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | 4.68 (10.74)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | 1.26 (4.35)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -0.06 (0.82)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | 0.23 (1.15)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -0.10 (1.27)
  Change at Month 72 of extension study: number analyzed (Participants) | 1
  Change at Month 72 of extension study | 2.80
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -0.40
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

52. Secondary Outcome: Change From Baseline (of Parent Study) in C-reactive Protein at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 50
Time Frame: Baseline of the parent study; Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milligram/Liter
Arm/Group | Etanercept
Number analyzed (Participants) | 13
milligram/Liter
  Change at Month 3 of extension study: number analyzed (Participants) | 11
  Change at Month 3 of extension study | -5.50 (11.59)
  Change at Month 6 of extension study | -5.99 (9.03)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -6.42 (9.72)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -6.91 (9.46)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -6.68 (8.88)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -7.79 (10.69)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -6.13 (11.41)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -5.18 (11.87)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | 2.76 (28.99)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | 0.60 (18.68)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | 0.22 (19.92)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | 20.44 (46.78)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -0.10 (0.58)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | 0.57 (2.54)
  Change at Month 78 of extension study: number analyzed (Participants) | 2
  Change at Month 78 of extension study | 5.30 (8.63)
  Change at Month 96 of extension study: number analyzed (Participants) | 0

53. Secondary Outcome: Change From Baseline (of Parent Study) in Visual Analogue Scale (VAS) Pain Score at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: VAS: 10-point pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. A higher score indicates greater pain intensity.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 15
  Change at Month 6 of extension study | -3.43 (2.05)
  Change at Month 12 of extension study: number analyzed (Participants) | 54
  Change at Month 12 of extension study | -4.02 (2.52)
  Change at Month 18 of extension study: number analyzed (Participants) | 64
  Change at Month 18 of extension study | -4.24 (2.58)
  Change at Month 24 of extension study: number analyzed (Participants) | 57
  Change at Month 24 of extension study | -4.40 (2.44)
  Change at Month 30 of extension study: number analyzed (Participants) | 58
  Change at Month 30 of extension study | -4.26 (2.50)
  Change at Month 36 of extension study: number analyzed (Participants) | 56
  Change at Month 36 of extension study | -4.03 (2.55)
  Change at Month 42 of extension study: number analyzed (Participants) | 50
  Change at Month 42 of extension study | -3.82 (3.21)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -4.15 (2.55)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -4.51 (2.65)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -4.36 (2.44)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -4.26 (2.67)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -4.19 (2.58)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -4.25 (2.17)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -4.09 (2.26)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -4.20 (2.60)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -4.39 (2.36)

54. Secondary Outcome: Change From Baseline (of Parent Study) in Visual Analogue Scale (VAS) Pain Score at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 53
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1 of extension study: number analyzed (Participants) | 22
  Change at Month 1 of extension study | -4.75 (2.79)
  Change at Month 3 of extension study: number analyzed (Participants) | 15
  Change at Month 3 of extension study | -4.03 (2.97)
  Change at Month 6 of extension study: number analyzed (Participants) | 11
  Change at Month 6 of extension study | -5.00 (2.66)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -4.36 (2.93)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -4.70 (2.80)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -4.50 (2.89)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -3.81 (2.49)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -3.36 (3.00)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -4.00 (2.93)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -3.67 (3.06)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -2.50 (3.54)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -3.67 (3.25)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -3.50 (3.50)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -3.75 (4.60)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -3.75 (4.60)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -0.50
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

55. Secondary Outcome: Change From Baseline (of Parent Study) in Visual Analogue Scale (VAS) Pain Score at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 53
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3 of extension study: number analyzed (Participants) | 11
  Change at Month 3 of extension study | -2.64 (2.68)
  Change at Month 6 of extension study | -2.65 (3.20)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -2.68 (2.92)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -3.05 (3.72)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -2.25 (3.23)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -2.25 (3.01)
  Change at Month 30 of extension study: number analyzed (Participants) | 8
  Change at Month 30 of extension study | -2.13 (3.06)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -2.29 (3.44)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -2.57 (3.05)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -1.75 (1.89)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -1.75 (2.12)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -0.90 (0.42)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -0.50 (0.71)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -0.83 (0.76)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | 0.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

56. Secondary Outcome: Change From Baseline (of Parent Study) in Duration of Morning Stiffness at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (if none was present = 0; if stiffness persisted the entire day = 1440 minutes was recorded; if morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported).
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Minutes
  Change at Month 6 of extension study: number analyzed (Participants) | 19
  Change at Month 6 of extension study | -52.11 (56.63)
  Change at Month 12 of extension study: number analyzed (Participants) | 57
  Change at Month 12 of extension study | -73.33 (110.91)
  Change at Month 18 of extension study: number analyzed (Participants) | 67
  Change at Month 18 of extension study | -80.24 (108.79)
  Change at Month 24 of extension study: number analyzed (Participants) | 63
  Change at Month 24 of extension study | -72.19 (105.84)
  Change at Month 30 of extension study: number analyzed (Participants) | 59
  Change at Month 30 of extension study | -66.36 (110.79)
  Change at Month 36 of extension study: number analyzed (Participants) | 56
  Change at Month 36 of extension study | -75.04 (112.27)
  Change at Month 42 of extension study: number analyzed (Participants) | 52
  Change at Month 42 of extension study | -73.75 (111.59)
  Change at Month 48 of extension study: number analyzed (Participants) | 49
  Change at Month 48 of extension study | -76.22 (118.95)
  Change at Month 54 of extension study: number analyzed (Participants) | 42
  Change at Month 54 of extension study | -82.21 (124.19)
  Change at Month 60 of extension study: number analyzed (Participants) | 39
  Change at Month 60 of extension study | -89.10 (126.62)
  Change at Month 66 of extension study: number analyzed (Participants) | 36
  Change at Month 66 of extension study | -95.56 (134.35)
  Change at Month 72 of extension study: number analyzed (Participants) | 34
  Change at Month 72 of extension study | -89.26 (148.76)
  Change at Month 78 of extension study: number analyzed (Participants) | 30
  Change at Month 78 of extension study | -91.17 (141.86)
  Change at Month 84 of extension study: number analyzed (Participants) | 29
  Change at Month 84 of extension study | -91.83 (143.82)
  Change at Month 90 of extension study: number analyzed (Participants) | 27
  Change at Month 90 of extension study | -101.85 (140.75)
  Change at Month 96 of extension study: number analyzed (Participants) | 23
  Change at Month 96 of extension study | -99.78 (152.26)

57. Secondary Outcome: Change From Baseline (of Parent Study) in Duration of Morning Stiffness at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (if none was present = 0; if stiffness persisted the entire day, 1440 minutes was recorded; if morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported).
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Minutes
  Change at Month 1 of extension study: number analyzed (Participants) | 23
  Change at Month 1 of extension study | -83.96 (119.42)
  Change at Month 3 of extension study: number analyzed (Participants) | 14
  Change at Month 3 of extension study | -71.43 (98.85)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -56.67 (62.32)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -29.09 (26.72)
  Change at Month 12 of extension study: number analyzed (Participants) | 10
  Change at Month 12 of extension study | -32.00 (26.27)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -32.00 (26.27)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -30.63 (29.33)
  Change at Month 30 of extension study: number analyzed (Participants) | 7
  Change at Month 30 of extension study | -30.71 (31.68)
  Change at Month 36 of extension study: number analyzed (Participants) | 7
  Change at Month 36 of extension study | -30.71 (31.68)
  Change at Month 42 of extension study: number analyzed (Participants) | 6
  Change at Month 42 of extension study | -25.83 (31.69)
  Change at Month 48 of extension study: number analyzed (Participants) | 4
  Change at Month 48 of extension study | -31.25 (37.50)
  Change at Month 54 of extension study: number analyzed (Participants) | 3
  Change at Month 54 of extension study | -41.67 (38.19)
  Change at Month 60 of extension study: number analyzed (Participants) | 3
  Change at Month 60 of extension study | -41.67 (38.19)
  Change at Month 66 of extension study: number analyzed (Participants) | 2
  Change at Month 66 of extension study | -25.00 (35.36)
  Change at Month 72 of extension study: number analyzed (Participants) | 2
  Change at Month 72 of extension study | -25.00 (35.36)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | 0.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

58. Secondary Outcome: Change From Baseline (of Parent Study) in Duration of Morning Stiffness at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 57
Time Frame: as for outcome 34
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Minutes
  Change at Month 3 of extension study | -116.15 (138.82)
  Change at Month 6 of extension study | -107.69 (147.90)
  Change at Month 9 of extension study: number analyzed (Participants) | 12
  Change at Month 9 of extension study | -126.67 (144.23)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -130.00 (151.53)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -111.00 (142.53)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -85.63 (137.98)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -72.22 (142.55)
  Change at Month 36 of extension study: number analyzed (Participants) | 8
  Change at Month 36 of extension study | -89.38 (135.24)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -101.43 (140.88)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -60.00 (94.45)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -60.00 (94.45)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -24.00 (37.82)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -7.50 (9.57)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -10.00 (10.00)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -20.00
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

59. Secondary Outcome: Percentage of Participants With Clinically Inactive Disease at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: Clinically inactive disease was defined as no joints with active arthritis; no fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA; no active uveitis; normal range of CRP; PGA of disease activity of 0 on a 21-circle VAS and duration of morning stiffness of less than or equal to (<=) 15 minutes.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of participants
  Month 6: number analyzed (Participants) | 68
  Month 6 | 11.8 [5.2 to 21.9]
  Month 12: number analyzed (Participants) | 70
  Month 12 | 25.7 [16.0 to 37.6]
  Month 18: number analyzed (Participants) | 69
  Month 18 | 36.2 [25.0 to 48.7]
  Month 24: number analyzed (Participants) | 62
  Month 24 | 24.2 [14.2 to 36.7]
  Month 30: number analyzed (Participants) | 59
  Month 30 | 30.5 [19.2 to 43.9]
  Month 36: number analyzed (Participants) | 56
  Month 36 | 32.1 [20.3 to 46.0]
  Month 42: number analyzed (Participants) | 53
  Month 42 | 32.1 [19.9 to 46.3]
  Month 48: number analyzed (Participants) | 49
  Month 48 | 28.6 [16.6 to 43.3]
  Month 54: number analyzed (Participants) | 42
  Month 54 | 33.3 [19.6 to 49.5]
  Month 60: number analyzed (Participants) | 39
  Month 60 | 30.8 [17.0 to 47.6]
  Month 66: number analyzed (Participants) | 36
  Month 66 | 25.0 [12.1 to 42.2]
  Month 72: number analyzed (Participants) | 33
  Month 72 | 12.1 [3.4 to 28.2]
  Month 78: number analyzed (Participants) | 30
  Month 78 | 23.3 [9.9 to 42.3]
  Month 84: number analyzed (Participants) | 29
  Month 84 | 27.6 [12.7 to 47.2]
  Month 90: number analyzed (Participants) | 27
  Month 90 | 25.9 [11.1 to 46.3]
  Month 96: number analyzed (Participants) | 23
  Month 96 | 26.1 [10.2 to 48.4]

60. Secondary Outcome: Percentage of Participants With Clinically Inactive Disease at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: Clinically inactive disease was defined as no joints with active arthritis; no fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA; no active uveitis; normal range of CRP; PGA of disease activity of 0 on a 21-circle VAS and duration of morning stiffness of <=15 minutes.
Time Frame: Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 withdrawal period of extension study
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Percentage of participants
  Month 1: number analyzed (Participants) | 22
  Month 1 | 54.5 [32.2 to 75.6]
  Month 3: number analyzed (Participants) | 15
  Month 3 | 66.7 [38.4 to 88.2]
  Month 6: number analyzed (Participants) | 12
  Month 6 | 66.7 [34.9 to 90.1]
  Month 9: number analyzed (Participants) | 11
  Month 9 | 81.8 [48.2 to 97.7]
  Month 12: number analyzed (Participants) | 10
  Month 12 | 80.0 [44.4 to 97.5]
  Month 18: number analyzed (Participants) | 10
  Month 18 | 80.0 [44.4 to 97.5]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 87.5 [47.3 to 99.7]
  Month 30: number analyzed (Participants) | 7
  Month 30 | 71.4 [29.0 to 96.3]
  Month 36: number analyzed (Participants) | 6
  Month 36 | 83.3 [35.9 to 99.6]
  Month 42: number analyzed (Participants) | 6
  Month 42 | 50.0 [11.8 to 88.2]
  Month 48: number analyzed (Participants) | 4
  Month 48 | 50.0 [6.8 to 93.2]
  Month 54: number analyzed (Participants) | 3
  Month 54 | 66.7 [9.4 to 99.2]
  Month 60: number analyzed (Participants) | 3
  Month 60 | 100 [29.2 to 100]
  Month 66: number analyzed (Participants) | 2
  Month 66 | 100 [15.8 to 100]
  Month 72: number analyzed (Participants) | 2
  Month 72 | 0.0 [0.0 to 84.2]
  Month 78: number analyzed (Participants) | 1
  Month 78 | 0.0 [0.0 to 97.5]
  Month 84: number analyzed (Participants) | 0
  Month 90: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

61. Secondary Outcome: Percentage of Participants With Clinically Inactive Disease at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 60
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 re-treatment period of extension study
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percentage of participants
  Month 3 | 23.1 [5.0 to 53.8]
  Month 6 | 46.2 [19.2 to 74.9]
  Month 9: number analyzed (Participants) | 12
  Month 9 | 33.3 [9.9 to 65.1]
  Month 12: number analyzed (Participants) | 11
  Month 12 | 45.5 [16.7 to 76.6]
  Month 18: number analyzed (Participants) | 10
  Month 18 | 50.0 [18.7 to 81.3]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 62.5 [24.5 to 91.5]
  Month 30: number analyzed (Participants) | 9
  Month 30 | 33.3 [7.5 to 70.1]
  Month 36: number analyzed (Participants) | 9
  Month 36 | 55.6 [21.2 to 86.3]
  Month 42: number analyzed (Participants) | 7
  Month 42 | 28.6 [3.7 to 71.0]
  Month 48: number analyzed (Participants) | 6
  Month 48 | 16.7 [0.4 to 64.1]
  Month 54: number analyzed (Participants) | 6
  Month 54 | 33.3 [4.3 to 77.7]
  Month 60: number analyzed (Participants) | 5
  Month 60 | 40.0 [5.3 to 85.3]
  Month 66: number analyzed (Participants) | 4
  Month 66 | 50.0 [6.8 to 93.2]
  Month 72: number analyzed (Participants) | 3
  Month 72 | 33.3 [0.8 to 90.6]
  Month 78: number analyzed (Participants) | 2
  Month 78 | 50.0 [1.3 to 98.7]
  Month 84: number analyzed (Participants) | 0
  Month 90: number analyzed (Participants) | 0
  Month 96: number analyzed (Participants) | 0

62. Secondary Outcome: Change From Baseline (of Parent Study) in Juvenile Arthritis Disease Activity Score 73 Joints (JADAS-73) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: JADAS-73 is a validated composite disease activity measure for JIA. It was derived from four components; 1) Physician global assessment of disease activity (assessed on 10 cm VAS, where 0= no activity and 10=maximum activity, higher scores indicated more disease activity). 2) Parent/participant global assessment of overall well-being (assessed on a VAS, where 0= very well and 10=very poor, higher scores indicated worse condition). 3) Number of joints with active disease (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness). 4) An inflammatory marker, CRP that was measured in mg/L and its value normalized to 0 to 10 scale, where higher scores indicated more disease activity. JADAS total score was calculated as the sum of its four components and ranged from 0-103. A higher score indicates more disease activity.
Time Frame: as for outcome 35
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 23
  Change at Month 6 of extension study | -15.00 (8.08)
  Change at Month 12 of extension study: number analyzed (Participants) | 57
  Change at Month 12 of extension study | -15.09 (8.01)
  Change at Month 18 of extension study: number analyzed (Participants) | 61
  Change at Month 18 of extension study | -15.83 (9.11)
  Change at Month 24 of extension study: number analyzed (Participants) | 59
  Change at Month 24 of extension study | -15.73 (7.84)
  Change at Month 30 of extension study: number analyzed (Participants) | 57
  Change at Month 30 of extension study | -15.54 (7.51)
  Change at Month 36 of extension study: number analyzed (Participants) | 50
  Change at Month 36 of extension study | -15.89 (7.40)
  Change at Month 42 of extension study: number analyzed (Participants) | 47
  Change at Month 42 of extension study | -16.23 (8.42)
  Change at Month 48 of extension study: number analyzed (Participants) | 46
  Change at Month 48 of extension study | -16.65 (7.70)
  Change at Month 54 of extension study: number analyzed (Participants) | 40
  Change at Month 54 of extension study | -17.68 (8.15)
  Change at Month 60 of extension study: number analyzed (Participants) | 36
  Change at Month 60 of extension study | -17.26 (6.90)
  Change at Month 66 of extension study: number analyzed (Participants) | 34
  Change at Month 66 of extension study | -17.19 (6.79)
  Change at Month 72 of extension study: number analyzed (Participants) | 30
  Change at Month 72 of extension study | -17.48 (6.77)
  Change at Month 78 of extension study: number analyzed (Participants) | 25
  Change at Month 78 of extension study | -17.13 (4.66)
  Change at Month 84 of extension study: number analyzed (Participants) | 26
  Change at Month 84 of extension study | -16.68 (4.81)
  Change at Month 90 of extension study: number analyzed (Participants) | 25
  Change at Month 90 of extension study | -17.18 (4.51)
  Change at Month 96 of extension study: number analyzed (Participants) | 21
  Change at Month 96 of extension study | -16.92 (4.75)

63. Secondary Outcome: Change From Baseline (of Parent Study) in Juvenile Arthritis Disease Activity Score 73 Joints (JADAS-73) Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period
Description: as for outcome 62
Time Frame: as for outcome 33
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 30
Units on scale
  Change at Month 1 of extension study: number analyzed (Participants) | 19
  Change at Month 1 of extension study | -16.66 (8.96)
  Change at Month 3 of extension study: number analyzed (Participants) | 14
  Change at Month 3 of extension study | -17.90 (9.04)
  Change at Month 6 of extension study: number analyzed (Participants) | 10
  Change at Month 6 of extension study | -20.41 (8.34)
  Change at Month 9 of extension study: number analyzed (Participants) | 8
  Change at Month 9 of extension study | -20.25 (9.45)
  Change at Month 12 of extension study: number analyzed (Participants) | 8
  Change at Month 12 of extension study | -20.19 (9.36)
  Change at Month 18 of extension study: number analyzed (Participants) | 8
  Change at Month 18 of extension study | -19.44 (9.83)
  Change at Month 24 of extension study: number analyzed (Participants) | 6
  Change at Month 24 of extension study | -19.42 (9.18)
  Change at Month 30 of extension study: number analyzed (Participants) | 5
  Change at Month 30 of extension study | -16.60 (6.32)
  Change at Month 36 of extension study: number analyzed (Participants) | 4
  Change at Month 36 of extension study | -15.50 (7.33)
  Change at Month 42 of extension study: number analyzed (Participants) | 5
  Change at Month 42 of extension study | -16.10 (6.58)
  Change at Month 48 of extension study: number analyzed (Participants) | 3
  Change at Month 48 of extension study | -17.83 (7.18)
  Change at Month 54 of extension study: number analyzed (Participants) | 2
  Change at Month 54 of extension study | -19.25 (9.55)
  Change at Month 60 of extension study: number analyzed (Participants) | 2
  Change at Month 60 of extension study | -19.50 (9.19)
  Change at Month 66 of extension study: number analyzed (Participants) | 1
  Change at Month 66 of extension study | -26.00
  Change at Month 72 of extension study: number analyzed (Participants) | 0
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

64. Secondary Outcome: Change From Baseline (of Parent Study) in Juvenile Arthritis Disease Activity Score 73 Joints (JADAS-73) at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period
Description: as for outcome 62
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 withdrawal period of extension study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Units on scale
  Change at Month 3 of extension study: number analyzed (Participants) | 11
  Change at Month 3 of extension study | -13.59 (6.06)
  Change at Month 6 of extension study: number analyzed (Participants) | 12
  Change at Month 6 of extension study | -13.80 (6.68)
  Change at Month 9 of extension study: number analyzed (Participants) | 11
  Change at Month 9 of extension study | -14.39 (7.98)
  Change at Month 12 of extension study: number analyzed (Participants) | 11
  Change at Month 12 of extension study | -13.26 (9.31)
  Change at Month 18 of extension study: number analyzed (Participants) | 10
  Change at Month 18 of extension study | -13.51 (8.78)
  Change at Month 24 of extension study: number analyzed (Participants) | 8
  Change at Month 24 of extension study | -12.68 (8.45)
  Change at Month 30 of extension study: number analyzed (Participants) | 9
  Change at Month 30 of extension study | -12.04 (7.89)
  Change at Month 36 of extension study: number analyzed (Participants) | 9
  Change at Month 36 of extension study | -12.90 (7.47)
  Change at Month 42 of extension study: number analyzed (Participants) | 7
  Change at Month 42 of extension study | -12.45 (9.24)
  Change at Month 48 of extension study: number analyzed (Participants) | 6
  Change at Month 48 of extension study | -10.85 (6.66)
  Change at Month 54 of extension study: number analyzed (Participants) | 6
  Change at Month 54 of extension study | -10.85 (5.96)
  Change at Month 60 of extension study: number analyzed (Participants) | 5
  Change at Month 60 of extension study | -6.82 (4.33)
  Change at Month 66 of extension study: number analyzed (Participants) | 4
  Change at Month 66 of extension study | -8.50 (2.12)
  Change at Month 72 of extension study: number analyzed (Participants) | 3
  Change at Month 72 of extension study | -8.17 (2.25)
  Change at Month 78 of extension study: number analyzed (Participants) | 1
  Change at Month 78 of extension study | -10.50
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

65. Secondary Outcome: Change From Baseline (of Parent Study) in Overall Back Pain at Month 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96 of Extension Study: Active Treatment Period: Enthesitis-Related Arthritis (ERA)
Description: Overall back pain assessed by participant's parent using a 100 millimeter (mm) VAS with 0 mm= no pain and 100 mm= most severe pain, higher scores indicated more pain.
Time Frame: Baseline of the parent study; Month 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: FAS included all participants in the parent study who received at least 1 dose of investigational product regardless of whether they received any investigational product during the extension study. Here, "Number of Participants Analyzed", signifies participants with ERA and "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 31
millimeter
  Change at Month 12 of extension study: number analyzed (Participants) | 21
  Change at Month 12 of extension study | -19.88 (27.66)
  Change at Month 18 of extension study: number analyzed (Participants) | 25
  Change at Month 18 of extension study | -21.66 (28.26)
  Change at Month 24 of extension study: number analyzed (Participants) | 22
  Change at Month 24 of extension study | -20.34 (30.98)
  Change at Month 30 of extension study: number analyzed (Participants) | 20
  Change at Month 30 of extension study | -20.08 (31.57)
  Change at Month 36 of extension study: number analyzed (Participants) | 20
  Change at Month 36 of extension study | -21.50 (28.70)
  Change at Month 42 of extension study: number analyzed (Participants) | 19
  Change at Month 42 of extension study | -21.69 (31.79)
  Change at Month 48 of extension study: number analyzed (Participants) | 18
  Change at Month 48 of extension study | -20.37 (34.06)
  Change at Month 54 of extension study: number analyzed (Participants) | 14
  Change at Month 54 of extension study | -20.98 (34.18)
  Change at Month 60 of extension study: number analyzed (Participants) | 12
  Change at Month 60 of extension study | -20.14 (25.00)
  Change at Month 66 of extension study: number analyzed (Participants) | 11
  Change at Month 66 of extension study | -18.15 (26.87)
  Change at Month 72 of extension study: number analyzed (Participants) | 11
  Change at Month 72 of extension study | -18.52 (24.80)
  Change at Month 78 of extension study: number analyzed (Participants) | 10
  Change at Month 78 of extension study | -16.07 (27.50)
  Change at Month 84 of extension study: number analyzed (Participants) | 10
  Change at Month 84 of extension study | -17.07 (28.19)
  Change at Month 90 of extension study: number analyzed (Participants) | 10
  Change at Month 90 of extension study | -17.57 (29.17)
  Change at Month 96 of extension study: number analyzed (Participants) | 8
  Change at Month 96 of extension study | -20.84 (30.08)

66. Secondary Outcome: Change From Baseline (of Parent Study) in Overall Back Pain at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period: Enthesitis-Related Arthritis (ERA)
Description: as for outcome 65
Time Frame: as for outcome 33
Population: WAS included participants who entered the withdrawal period. Here, "Number of Participants Analyzed", signifies participants with ERA and "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 9
millimeter
  Change at Month 1 of extension study: number analyzed (Participants) | 7
  Change at Month 1 of extension study | -18.13 (26.75)
  Change at Month 3 of extension study: number analyzed (Participants) | 4
  Change at Month 3 of extension study | -27.48 (33.22)
  Change at Month 6 of extension study: number analyzed (Participants) | 3
  Change at Month 6 of extension study | -35.21 (33.07)
  Change at Month 9 of extension study: number analyzed (Participants) | 2
  Change at Month 9 of extension study | -30.50 (51.62)
  Change at Month 12 of extension study: number analyzed (Participants) | 2
  Change at Month 12 of extension study | -32.00 (49.50)
  Change at Month 18 of extension study: number analyzed (Participants) | 2
  Change at Month 18 of extension study | -33.50 (47.38)
  Change at Month 24 of extension study: number analyzed (Participants) | 2
  Change at Month 24 of extension study | -33.50 (47.38)
  Change at Month 30 of extension study: number analyzed (Participants) | 2
  Change at Month 30 of extension study | -14.00 (74.95)
  Change at Month 36 of extension study: number analyzed (Participants) | 2
  Change at Month 36 of extension study | -29.00 (53.74)
  Change at Month 42 of extension study: number analyzed (Participants) | 2
  Change at Month 42 of extension study | -34.00 (46.67)
  Change at Month 48 of extension study: number analyzed (Participants) | 0
  Change at Month 54 of extension study: number analyzed (Participants) | 0
  Change at Month 60 of extension study: number analyzed (Participants) | 0
  Change at Month 66 of extension study: number analyzed (Participants) | 0
  Change at Month 72 of extension study: number analyzed (Participants) | 0
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

67. Secondary Outcome: Change From Baseline (of Parent Study) in Overall Back Pain at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period: Enthesitis-Related Arthritis (ERA)
Description: Overall back pain assessed by participant's parent using a 100 mm VAS with 0 mm= no pain and 100 mm= most severe pain, higher scores indicated more pain.
Time Frame: as for outcome 34
Population: RTAS included those participants who entered the re-treatment period. Here, "Number of Participants Analyzed", signifies participants with ERA and "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 2
millimeter
  Change at Month 3 of extension study | -21.00 (7.07)
  Change at Month 6 of extension study | -29.00 (18.38)
  Change at Month 9 of extension study | -24.50 (12.02)
  Change at Month 12 of extension study | -23.50 (10.61)
  Change at Month 18 of extension study: number analyzed (Participants) | 1
  Change at Month 18 of extension study | -31.00
  Change at Month 30 of extension study: number analyzed (Participants) | 1
  Change at Month 30 of extension study | -13.00
  Change at Month 36 of extension study: number analyzed (Participants) | 1
  Change at Month 36 of extension study | -22.00
  Change at Month 42 of extension study: number analyzed (Participants) | 1
  Change at Month 42 of extension study | -26.00
  Change at Month 46 of extension study: number analyzed (Participants) | 1
  Change at Month 46 of extension study | -21.00
  Change at Month 54 of extension study: number analyzed (Participants) | 1
  Change at Month 54 of extension study | -26.00
  Change at Month 60 of extension study: number analyzed (Participants) | 1
  Change at Month 60 of extension study | -14.00
  Change at Month 66 of extension study: number analyzed (Participants) | 0
  Change at Month 72 of extension study: number analyzed (Participants) | 0
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

68. Secondary Outcome: Change From Baseline (of Parent Study) in Nocturnal Back Pain at Month 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96 of Extension Study: Active Treatment Period: Enthesitis-Related Arthritis (ERA)
Description: Nocturnal back pain assessed by participant's parent using a 100 mm VAS with 0 mm = no pain and 100 mm = most severe pain, higher scores indicated more pain.
Time Frame: as for outcome 65
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 31
millimeter
  Change at Month 12 of extension study: number analyzed (Participants) | 21
  Change at Month 12 of extension study | -17.41 (29.79)
  Change at Month 18 of extension study: number analyzed (Participants) | 25
  Change at Month 18 of extension study | -14.99 (28.13)
  Change at Month 24 of extension study: number analyzed (Participants) | 22
  Change at Month 24 of extension study | -16.90 (29.53)
  Change at Month 30 of extension study: number analyzed (Participants) | 20
  Change at Month 30 of extension study | -18.09 (31.21)
  Change at Month 36 of extension study: number analyzed (Participants) | 20
  Change at Month 36 of extension study | -17.31 (29.73)
  Change at Month 42 of extension study: number analyzed (Participants) | 19
  Change at Month 42 of extension study | -19.23 (30.56)
  Change at Month 48 of extension study: number analyzed (Participants) | 18
  Change at Month 48 of extension study | -19.16 (31.13)
  Change at Month 54 of extension study: number analyzed (Participants) | 14
  Change at Month 54 of extension study | -23.78 (33.66)
  Change at Month 60 of extension study: number analyzed (Participants) | 12
  Change at Month 60 of extension study | -19.83 (30.43)
  Change at Month 66 of extension study: number analyzed (Participants) | 11
  Change at Month 66 of extension study | -19.99 (29.90)
  Change at Month 72 of extension study: number analyzed (Participants) | 11
  Change at Month 72 of extension study | -16.45 (29.24)
  Change at Month 78 of extension study: number analyzed (Participants) | 10
  Change at Month 78 of extension study | -15.89 (30.10)
  Change at Month 84 of extension study: number analyzed (Participants) | 10
  Change at Month 84 of extension study | -18.49 (34.10)
  Change at Month 90 of extension study: number analyzed (Participants) | 10
  Change at Month 90 of extension study | -17.39 (37.42)
  Change at Month 96 of extension study: number analyzed (Participants) | 8
  Change at Month 96 of extension study | -22.49 (37.77)

69. Secondary Outcome: Change From Baseline (of Parent Study) in Nocturnal Back Pain at Month 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Withdrawal Period: Enthesitis-Related Arthritis (ERA)
Description: as for outcome 68
Time Frame: as for outcome 33
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 9
millimeter
  Change at Month 1 of extension study: number analyzed (Participants) | 7
  Change at Month 1 of extension study | -1.28 (3.45)
  Change at Month 3 of extension study: number analyzed (Participants) | 4
  Change at Month 3 of extension study | 0.02 (0.03)
  Change at Month 6 of extension study: number analyzed (Participants) | 3
  Change at Month 6 of extension study | 0.04 (1.06)
  Change at Month 9 of extension study: number analyzed (Participants) | 2
  Change at Month 9 of extension study | 0.50 (0.71)
  Change at Month 12 of extension study: number analyzed (Participants) | 2
  Change at Month 12 of extension study | -0.50 (0.71)
  Change at Month 18 of extension study: number analyzed (Participants) | 2
  Change at Month 18 of extension study | 0.00 (0.00)
  Change at Month 24 of extension study: number analyzed (Participants) | 2
  Change at Month 24 of extension study | 0.00 (0.00)
  Change at Month 30 of extension study: number analyzed (Participants) | 2
  Change at Month 30 of extension study | 11.50 (16.26)
  Change at Month 36 of extension study: number analyzed (Participants) | 2
  Change at Month 36 of extension study | 0.00 (0.00)
  Change at Month 42 of extension study: number analyzed (Participants) | 2
  Change at Month 42 of extension study | 0.00 (0.00)
  Change at Month 48 of extension study: number analyzed (Participants) | 0
  Change at Month 54 of extension study: number analyzed (Participants) | 0
  Change at Month 60 of extension study: number analyzed (Participants) | 0
  Change at Month 66 of extension study: number analyzed (Participants) | 0
  Change at Month 72 of extension study: number analyzed (Participants) | 0
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

70. Secondary Outcome: Change From Baseline (of Parent Study) in Nocturnal Back Pain at Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Re-treatment Period: Enthesitis-Related Arthritis (ERA)
Description: as for outcome 68
Time Frame: as for outcome 34
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Etanercept
Number analyzed (Participants) | 2
millimeter
  Change at Month 3 of extension study | -3.00 (8.49)
  Change at Month 6 of extension study | -6.00 (4.24)
  Change at Month 9 of extension study | -0.50 (12.02)
  Change at Month 12 of extension study | 0.00 (12.73)
  Change at Month 18 of extension study: number analyzed (Participants) | 1
  Change at Month 18 of extension study | 4.00
  Change at Month 30 of extension study: number analyzed (Participants) | 1
  Change at Month 30 of extension study | 14.00
  Change at Month 36 of extension study: number analyzed (Participants) | 1
  Change at Month 36 of extension study | 17.00
  Change at Month 42 of extension study: number analyzed (Participants) | 1
  Change at Month 42 of extension study | 7.00
  Change at Month 48 of extension study: number analyzed (Participants) | 1
  Change at Month 48 of extension study | 10.00
  Change at Month 54 of extension study: number analyzed (Participants) | 1
  Change at Month 54 of extension study | 5.00
  Change at Month 60 of extension study: number analyzed (Participants) | 1
  Change at Month 60 of extension study | 38.00
  Change at Month 66 of extension study: number analyzed (Participants) | 0
  Change at Month 72 of extension study: number analyzed (Participants) | 0
  Change at Month 78 of extension study: number analyzed (Participants) | 0
  Change at Month 84 of extension study: number analyzed (Participants) | 0
  Change at Month 90 of extension study: number analyzed (Participants) | 0
  Change at Month 96 of extension study: number analyzed (Participants) | 0

71. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Score at Month 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period: Enthesitis-Related Arthritis (ERA)
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored on a 3-point scale ranged from 0 to 2 (0=normal mobility, 2=severe reduction, where higher scores indicated more reduction). The total BASMI score range from 0 to 10, where higher scores indicated more reduction in spinal mobility.
Time Frame: Month 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 31
Units on scale
  Month 12: number analyzed (Participants) | 20
  Month 12 | 0.39 (0.64)
  Month 18: number analyzed (Participants) | 24
  Month 18 | 0.21 (0.51)
  Month 24: number analyzed (Participants) | 22
  Month 24 | 0.23 (0.53)
  Month 30: number analyzed (Participants) | 20
  Month 30 | 0.40 (0.68)
  Month 36: number analyzed (Participants) | 20
  Month 36 | 0.30 (0.66)
  Month 42: number analyzed (Participants) | 18
  Month 42 | 0.17 (0.51)
  Month 48: number analyzed (Participants) | 18
  Month 48 | 0.28 (0.67)
  Month 54: number analyzed (Participants) | 14
  Month 54 | 0.21 (0.58)
  Month 60: number analyzed (Participants) | 12
  Month 60 | 0.17 (0.39)
  Month 66: number analyzed (Participants) | 11
  Month 66 | 0.09 (0.30)
  Month 72: number analyzed (Participants) | 11
  Month 72 | 0.09 (0.30)
  Month 78: number analyzed (Participants) | 10
  Month 78 | 0.10 (0.32)
  Month 84: number analyzed (Participants) | 10
  Month 84 | 0.10 (0.32)
  Month 90: number analyzed (Participants) | 10
  Month 90 | 0.10 (0.32)
  Month 96: number analyzed (Participants) | 8
  Month 96 | 0.00 (0.00)

72. Secondary Outcome: Change From Baseline (of Parent Study) in Percentage Body Surface Area (BSA) at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period: Psoriatic Arthritis (PsA)
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method: one of the participant's palm to proximal interphalangeal and thumb= 1% of BSA. Regions of the body were assigned specific number of palms with percentage (Head and neck= 10% [10 palms], upper extremities= 20% [20 palms], Trunk [axillae and groin]= 30% [30 palms], lower extremities [buttocks]= 40% [40 palms]). The total BSA affected was the summation of individual regions affected.
Time Frame: as for outcome 35
Population: FAS included all participants in the parent study who received at least 1 dose of investigational product regardless of whether they received any investigational product during the extension study. Here, "Number of Participants Analyzed", signifies participants with PsA and "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | Etanercept
Number analyzed (Participants) | 23
Percentage of body surface area
  Change at Month 6 of extension study: number analyzed (Participants) | 10
  Change at Month 6 of extension study | -5.45 (10.36)
  Change at Month 12 of extension study: number analyzed (Participants) | 15
  Change at Month 12 of extension study | -10.07 (13.96)
  Change at Month 18 of extension study: number analyzed (Participants) | 15
  Change at Month 18 of extension study | -9.82 (12.55)
  Change at Month 24 of extension study: number analyzed (Participants) | 13
  Change at Month 24 of extension study | -11.85 (13.71)
  Change at Month 30 of extension study: number analyzed (Participants) | 14
  Change at Month 30 of extension study | -10.95 (14.42)
  Change at Month 36 of extension study: number analyzed (Participants) | 13
  Change at Month 36 of extension study | -10.38 (15.93)
  Change at Month 42 of extension study: number analyzed (Participants) | 14
  Change at Month 42 of extension study | -11.18 (14.21)
  Change at Month 48 of extension study: number analyzed (Participants) | 12
  Change at Month 48 of extension study | -11.81 (14.06)
  Change at Month 54 of extension study: number analyzed (Participants) | 11
  Change at Month 54 of extension study | -12.45 (14.34)
  Change at Month 60 of extension study: number analyzed (Participants) | 11
  Change at Month 60 of extension study | -12.09 (13.66)
  Change at Month 66 of extension study: number analyzed (Participants) | 10
  Change at Month 66 of extension study | -10.88 (13.38)
  Change at Month 72 of extension study: number analyzed (Participants) | 9
  Change at Month 72 of extension study | -8.88 (19.95)
  Change at Month 78 of extension study: number analyzed (Participants) | 8
  Change at Month 78 of extension study | -13.39 (14.64)
  Change at Month 84 of extension study: number analyzed (Participants) | 8
  Change at Month 84 of extension study | -13.50 (14.93)
  Change at Month 90 of extension study: number analyzed (Participants) | 6
  Change at Month 90 of extension study | -16.83 (15.83)
  Change at Month 96 of extension study: number analyzed (Participants) | 5
  Change at Month 96 of extension study | -15.80 (17.47)

73. Secondary Outcome: Change From Baseline (of Parent Study) in Physician's Global Assessment (PGA) of Psoriasis Score at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period: Psoriatic Arthritis (PsA)
Description: PGA of Psoriasis assessed the amount of induration, erythema, and scaling averaged over all psoriatic lesions on a scale of 0 to 5, where 0= no psoriasis to 5= severe disease, where higher scores indicated more severity. 'Clear' and "Almost clear' includes all participants who were scored as a 0 or 1.
Time Frame: as for outcome 35
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept
Number analyzed (Participants) | 23
Units on scale
  Change at Month 6 of extension study: number analyzed (Participants) | 9
  Change at Month 6 of extension study | -1.33 (1.41)
  Change at Month 12 of extension study: number analyzed (Participants) | 15
  Change at Month 12 of extension study | -1.33 (1.23)
  Change at Month 18 of extension study: number analyzed (Participants) | 15
  Change at Month 18 of extension study | -1.20 (1.26)
  Change at Month 24 of extension study: number analyzed (Participants) | 13
  Change at Month 24 of extension study | -1.54 (1.27)
  Change at Month 30 of extension study: number analyzed (Participants) | 14
  Change at Month 30 of extension study | -1.07 (1.49)
  Change at Month 36 of extension study: number analyzed (Participants) | 14
  Change at Month 36 of extension study | -1.21 (1.12)
  Change at Month 42 of extension study: number analyzed (Participants) | 14
  Change at Month 42 of extension study | -1.50 (1.22)
  Change at Month 48 of extension study: number analyzed (Participants) | 12
  Change at Month 48 of extension study | -1.42 (1.08)
  Change at Month 54 of extension study: number analyzed (Participants) | 11
  Change at Month 54 of extension study | -1.18 (1.33)
  Change at Month 60 of extension study: number analyzed (Participants) | 11
  Change at Month 60 of extension study | -1.18 (1.17)
  Change at Month 66 of extension study: number analyzed (Participants) | 10
  Change at Month 66 of extension study | -1.20 (0.92)
  Change at Month 72 of extension study: number analyzed (Participants) | 9
  Change at Month 72 of extension study | -1.11 (1.05)
  Change at Month 78 of extension study: number analyzed (Participants) | 8
  Change at Month 78 of extension study | -1.13 (1.13)
  Change at Month 84 of extension study: number analyzed (Participants) | 8
  Change at Month 84 of extension study | -1.50 (1.07)
  Change at Month 90 of extension study: number analyzed (Participants) | 6
  Change at Month 90 of extension study | -1.50 (1.05)
  Change at Month 96 of extension study: number analyzed (Participants) | 5
  Change at Month 96 of extension study | -1.80 (1.10)

74. Secondary Outcome: All Cause Mortality: All Periods of Extension Study
Description: The considered event was death due to any cause from baseline to the end of the study.
Time Frame: Extension study: First dose of study medication up to 30 days after last dose of study drug (maximum up to 97 months)
Population: The analysis set included all participants enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants | 0

75. Secondary Outcome: Number of Participants With Prior Non-study Medication: All Periods of Extension Study
Description: Prior non-study medications were defined as any non-study medications taken before the first dose of investigational product taken at the start of the study. These included anti-infective, corticosteroids, oral corticosteroids, Parenteral corticosteroids, disease-modifying antirheumatic drugs and oral non-steroidal anti-inflammatory medication.
Time Frame: Extension study: First dose of study medication up to 30 days after last dose of study drug (maximum up to 97 months)
Population: The analysis set included all participants enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants
  Anti-infective | 2
  Corticosteroids | 5
  Oral Corticosteroids | 5
  Parenteral Corticosteroid | 0
  Disease-modifying Antirheumatic Drugs | 57
  Oral Non-steroidal Anti-inflammatory Medication | 13

76. Secondary Outcome: Number of Participants With Concomitant Non-study Medication: All Periods of Extension Study
Description: Concomitant non-study medications were defined as any non-study medications taken during the treatment period. These included anti-infective medications, corticosteroids, oral corticosteroids, Parenteral corticosteroids, disease-modifying antirheumatic drugs, oral non-steroidal anti-inflammatory drugs and non-steroidal anti-inflammatory drugs.
Time Frame: Extension study: First dose of study medication up to 30 days after last dose of study drug (maximum up to 97 months)
Population: The analysis set included all participants enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants
  Anti-infective Medications | 62
  Corticosteroids | 29
  Oral Corticosteroids | 16
  Parenteral Corticosteroid | 12
  Disease-modifying Antirheumatic Drugs | 64
  Non-steroidal Anti-inflammatory Drugs | 51
  Oral Non-steroidal Anti-inflammatory Drugs | 48

77. Secondary Outcome: Number of Participants With After Non-study Medication: All Periods of Extension Study
Description: After non-study medications referred to any non-study medications taken after the last dose of the investigational product. These included anti-infective, corticosteroids, oral corticosteroids, Parenteral corticosteroids, disease-modifying antirheumatic drugs, oral non-steroidal anti-inflammatory medication and non-steroidal anti-inflammatory medication.
Time Frame: Extension study: Last dose of study medication up to 30 days (maximum up to 97 months)
Population: The analysis set included all participants enrolled in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 109
Participants
  Anti-infectives | 7
  Corticosteroids | 6
  Oral Corticosteroids | 3
  Parenteral Corticosteroid | 1
  Disease-modifying Antirheumatic Drugs | 48
  Non-steroidal Anti-inflammatory Drugs | 16
  Oral Non-steroidal Anti-inflammatory Drugs | 16

78. Secondary Outcome: Exposure Time: Extension Study: Active Treatment Period
Description: The exposure time (in years) to etanercept was calculated for each participant using the following formula: (the last dose date minus the first dose date plus 1)/365.25. If the gap was less than 28 days between two etanercept treatment periods, the cumulative exposure included the gap. Else, the gap was excluded from the cumulative exposure. Exposure time in year was converted into weeks and reported here.
Time Frame: Extension study: First dose of study medication up to 30 days after last dose of study drug (maximum up to 97 months)
Population: FAS included all participants in the parent study who received at least 1 dose of investigational product regardless of whether they received any investigational product during the extension study.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Weeks | 244.79 (147.71) [lower limit 147.71]

79. Secondary Outcome: Percentage of Participants With Total Childhood Health Assessment Questionnaire (CHAQ) Score Improvement of >0.188 at Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 of Extension Study: Active Treatment Period
Description: as for outcome 38
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 active treatment period of extension study
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Percentage of Participants
  Baseline: number analyzed (Participants) | 80
  Baseline | 68.8 [57.4 to 78.7]
  Month 6: number analyzed (Participants) | 74
  Month 6 | 73.0 [61.4 to 82.6]
  Month 12: number analyzed (Participants) | 62
  Month 12 | 79.0 [66.8 to 88.3]
  Month 18: number analyzed (Participants) | 46
  Month 18 | 78.3 [63.6 to 89.1]
  Month 24: number analyzed (Participants) | 37
  Month 24 | 86.5 [71.2 to 95.5]
  Month 30: number analyzed (Participants) | 32
  Month 30 | 90.6 [75.0 to 98.0]
  Month 36: number analyzed (Participants) | 22
  Month 36 | 90.9 [70.8 to 98.9]
  Month 42: number analyzed (Participants) | 21
  Month 42 | 95.2 [76.2 to 99.9]
  Month 48: number analyzed (Participants) | 16
  Month 48 | 93.8 [69.8 to 99.8]
  Month 54: number analyzed (Participants) | 10
  Month 54 | 100.0 [69.2 to 100.0]
  Month 60: number analyzed (Participants) | 8
  Month 60 | 100.0 [63.1 to 100.0]
  Month 66: number analyzed (Participants) | 7
  Month 66 | 100.0 [59.0 to 100.0]
  Month 72: number analyzed (Participants) | 6
  Month 72 | 100.0 [54.1 to 100.0]
  Month 78: number analyzed (Participants) | 5
  Month 78 | 100.0 [47.8 to 100.0]
  Month 84: number analyzed (Participants) | 4
  Month 84 | 100.0 [39.8 to 100.0]
  Month 90: number analyzed (Participants) | 4
  Month 90 | 100.0 [39.8 to 100.0]
  Month 96: number analyzed (Participants) | 2
  Month 96 | 100.0 [15.8 to 100.0]

80. Secondary Outcome: Number of Participants With Vital Signs Abnormalities: Extension Study: Active Treatment Period
Description: Vital signs assessment included temperature, pulse, systolic and diastolic blood pressure. Pulse rate was obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Month 96 active treatment period of extension study
Population: as for outcome 78
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 99
Participants
  Pulse (low) | 1
  Systolic blood pressure (high) | 14
  Diastolic blood pressure (low) | 4
  Diastolic blood pressure (high) | 2
  Temperature | 0

ADVERSE EVENTS:
Time Frame: Extension study: First dose of study medication up to 30 days after last dose of study drug (maximum up to 97 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study. AEs and SAEs were analysed for full analysis set.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/109
Serious Adverse Events (participants affected / at risk) | 22/109
Other Adverse Events (participants affected / at risk) | 85/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=109)
Iridocyclitis (Eye disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 2
Uveitis (Eye disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Varicocele (Reproductive system and breast disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Knee operation (Surgical and medical procedures) | 1
Varicose vein (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=109)
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Eustachian tube disorder (Ear and labyrinth disorders) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Iridocyclitis (Eye disorders) | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Maculopathy (Eye disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Uveitis (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 4
Aphthous ulcer (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Enteritis (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Pneumoperitoneum (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 2
Injection site reaction (General disorders) | 6
Pyrexia (General disorders) | 6
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 2
Peripheral swelling (General disorders) | 1
Acarodermatitis (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 4
Diarrhoea infectious (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 12
Ear infection (Infections and infestations) | 5
Enterovirus infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastrointestinal viral infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 8
Laryngitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 8
Oral herpes (Infections and infestations) | 2
Orchitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 3
Otitis media acute (Infections and infestations) | 1
Paronychia (Infections and infestations) | 3
Periodontitis (Infections and infestations) | 3
Pertussis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 21
Pharyngotonsillitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Pulpitis dental (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Respiratory tract infection viral (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 8
Staphylococcal skin infection (Infections and infestations) | 1
Suspected COVID-19 (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 28
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 3
Viraemia (Infections and infestations) | 1
Viral infection (Infections and infestations) | 4
Viral tonsillitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Facial bones fracture (Injury, poisoning and procedural complications) | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 2
Hand fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 4
Limb injury (Injury, poisoning and procedural complications) | 2
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Blood pressure increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Transaminases increased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Gastroenteritis (Infections and infestations) | 10
Gastroenteritis viral (Infections and infestations) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Herpes simplex (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Patella fracture (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2
Weight increased (Investigations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 3
Joint laxity (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 4
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 3
Acne conglobata (Skin and subcutaneous tissue disorders) | 1
Acne cystic (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Narcolepsy (Nervous system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT01421069/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT01421069/SAP_001.pdf